# CD34-Selected Allogeneic Hematopoietic Cell Transplantation with Myeloablative Conditioning and CD8<sup>+</sup> Memory T-cell Infusion For Patients with Myelodysplastic Syndrome, Acute Leukemia, and Chronic Myelogenous Leukemia

#### **Coordinating Center**

Stanford Cancer Center 875 Blake Wilbur Dr Stanford, CA 94305

#### **Protocol Director**

Robert Lowsky, MD
Division of Blood and Marrow Transplantation
Stanford University Medical Center
300 Pasteur Dr, Room H0101B, Stanford, CA 94305
650-723-0822; 650-725-8950
rlowsky@stanford.edu

IRB-49023 OnCore-BMT339 NCT04151706 IND 014844

Version date: 12 February 2021 SRC approval: 28 May 2019

#### **Co-Investigators**

IRB-49023 Page 1 of 43 12 February 2021 v4

#### **Co-Investigators**

Wen-Kai-Weng, MD, PhD
Division of Blood and Marrow Transplantation
Stanford University Medical Center
300 Pasteur Dr MC5623, Stanford, CA 94305
650-723-0822; 650-725-8950
wkweng@stanford.edu

Robert Negrin, MD
Division of Blood and Marrow Transplantation
Stanford University Medical Center
300 Pasteur Dr MC5623, Stanford, CA 94305
650-723-0822; 650-725-8950
negrs@stanford.edu

Sally Arai, MD
Division of Blood and Marrow Transplantation
Stanford University Medical Center
300 Pasteur Dr MC5623, Stanford, CA 94305
650-723-0822; 650-725-8950
sarai1@stanford.edu

Laura Johnston, MD

Division of Blood and Marrow Transplantation
Stanford University Medical Center
300 Pasteur Dr MC5623, Stanford, CA 94305
650-723-0822; 650-725-8950
korb@stanford.edu

#### **Co-Investigators**

David Miklos, MD, PhD
Division of Blood and Marrow Transplantation
Stanford University Medical Center
300 Pasteur Dr MC5623, Stanford, CA 94305
650-723-0822; 650-725-8950
dmiklos@stanford.edu

Judith Shizuru, MD, PhD
Division of Blood and Marrow Transplantation
Stanford University Medical Center
300 Pasteur Dr MC5623, Stanford, CA 94305
650-723-0822; 650-725-8950
Jshizuru@stanford.edu

Everett Meyer, MD, PhD

Division of Blood and Marrow Transplantation
and Cellular Therapeutics Facility Laboratory
Stanford University Medical Center
300 Pasteur Dr MC5623, Stanford, CA 94305
650-723-0822; 650-725-8950
evmeyer@stanford.edu

Andrew Rezvani, MD

Division of Blood and Marrow Transplantation
Stanford University Medical Center
300 Pasteur Dr MC5623, Stanford, CA 94305
650-723-0822; 650-725-8950
arezvani@stanford.edu

Lori Muffly, MD

Division of Blood and Marrow Transplantation
Stanford University Medical Center
300 Pasteur Dr MC5623, Stanford, CA 94305
650-723-0822; 650-725-8950
lmuffly@stanford.edu

Samuel Strober, MD
Divisions of Immunology & Rheumatology
CCSR Building, Room 2215-C
Stanford, California 94305
650-723-6500; 650-725-6104
sstrober@stanford.edu

Michael Spinner, MD

Division of Blood and Marrow Transplantation
Stanford University Medical Center

300 Pasteur Drive MC5623, Stanford, CA 94305
650-723-0822; 650-725-8950
mspinner@stanford.edu

Parveen Shiraz, MD
Division of Blood and Marrow Transplantation
Stanford University Medical Center
300 Pasteur Dr MC5623, Stanford, CA 94305
650-723-0820; 650-725-8950
pshiraz@stanford.edu

Surbhi Sidana, MD
Division of Blood and Marrow Transplantation
Stanford University Medical Center
300 Pasteur Dr MC5623, Stanford, CA 94305
650-723-1389; 650-725-8950
surbhi.sidana@stanford.edu

Philip Lavori, PhD (Biostatistician)
Department of Health Research and Policy
Biostatistics Shared Resource,
Redwood Building, T101E, Stanford, CA 94305
650-725-6109; 650-725-6951
lavori@stanford.edu

#### **TABLE OF CONTENTS**

| Prote | ocol Synopsis | 4 |
|-------|------------------------------------------------|----|
| Prote | ocol Schema | 5 |
| 1. | Objectives | 6 |
| 2. | Background | 8 |
| 3. | Participant Selection and Eligibility Criteria | 20 |
| 4. | Treatment Plan | 27 |
| 5. | Investigational Agent Information | 29 |
| 6. | Dose Modification | 30 |
| 7. | Adverse Events and Reporting Procedures | 30 |
| 8. | Correlative Studies | 31 |
| 9. | Study Calendar | 32 |
| 10. | Measurements | 32 |
| 11. | Regulatory Considerations | 33 |
| 12. | Statistical Considerations | 34 |
| 13. | References | 36 |
| Appe | endices | 40 |

#### **Protocol Synopsis**

| TITLE | CD34-selected allogeneic hematopoietic cell transplantation with myeloablative conditioning and CD8 <sup>+</sup> memory T-cell infusion for patients with myelodysplastic syndrome, acute leukemia, and chronic myelogenous leukemia (CML) |
|---|---|
| STUDY PHASE | Phase 2 |
| STUDY DESIGN | Single-arm, non-randomized safety and efficacy study using Simon stage 2 design |
| STUDY SITE | Stanford University Medical Center, CA 94305 |
| INDICATION | Subjects with myelodysplastic syndrome (MDS), acute myeloid leukemia (AML), or acute lymphoblastic leukemia (ALL) eligible for full-dose myeloablative conditioning, or chronic myelogenous leukemia (CML) |
| INVESTIGATIONAL PRODUCT | Allogeneic phenotypic CD8 <sup>+</sup> memory T-cells from HLA-matched donors infused at the time of hematopoietic cell transplantation |
| PRIMARY ENDPOINT and OBJECTIVE(S) | To determine the rate of graft-versus-host-disease (GvHD)-free, relapse-free survival (GRFS) at one year post-transplant |
| SECONDARY<br>ENDPOINTS AND<br>OBJECTIVE(S) | To determine the rate of graft rejection, acute and chronic GvHD, non-relapse mortality, relapse, overall survival, disease-free survival, EBV and CMV reactivation, and the expansion and migration of EBV and CMV-reactive CD8 <sup>+</sup> memory T-cells |
| STUDY<br>OBSERVATION<br>PERIOD | The total duration of subject study participation is 1 year. Subjects will be followed indefinitely for all outcomes including overall survival, disease-free survival, and late complications including chronic GvHD and infections. |
| TREATMENT<br>SUMMARY | CD34 selection with immunomagnetic beads is an effective method of depleting alloreactive donor T-cells from a peripheral blood graft and results in a significant reduction in acute and chronic GvHD. However, depletion of donor T-cells also leads to an increased rate of disease relapse and infection. We will test the hypothesis that combining phenotypic CD8 <sup>+</sup> memory T-cells to a purified CD34 <sup>+</sup> graft will retain the low incidence of GvHD, yet also provide enhanced antitumor activity, and transfer of EBV and CMV immunity. |
| SAMPLE SIZE | 32 subjects and HLA-matched donors. |

| SUMMARY OF<br>SUBJECT<br>ELIGIBILTY | Subjects with histologically-confirmed MDS, acute leukemia, or CML. Subjects age 18 to 65 years who are eligible for full-dose myeloablative conditioning. Subjects with HLA-matched donors. |
|---|---|
| CONTROL GROUP | Historically-matched control subjects with MDS, AML, ALL, or CML receiving CD34-selected transplants with myeloablative conditioning without CD8 <sup>+</sup> memory T-cell infusion |

#### **Study Schema**



Donors will undergo apheresis for processing of CD34<sup>+</sup> selected cells and CD8<sup>+</sup>CD45RA<sup>-</sup> T<sub>M</sub> cells. These cells will be infused on Day 0 following a standard non-ATG containing regimen used for CD34-selected transplants consisting of fTBI (1375 cGy); thiotepa (10 mg/kg); and fludarabine (125 mg/m<sup>2</sup>) or non-TBI conditioning consisting of Busulfan (14.4 mg/kg) and Cyclophosphamide (120 mg/kg).

#### 1. OBJECTIVES

#### 1.1 Objectives

#### 1.1.1 Primary Objective

To determine the rate of graft-versus-host-disease (GvHD)-free, relapse-free survival (GRFS) at one year following CD34-selected allogeneic hematopoietic cell transplantation using myeloablative conditioning combined with an infusion of phenotypic CD8<sup>+</sup> memory T-cells from HLA-matched donors for subjects with myelodysplastic syndrome (MDS), acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), or chronic myelogenous leukemia (CML).

#### 1.1.2 Secondary Objectives

To determine the rate of graft rejection, acute and chronic GvHD, non-relapse mortality, relapse, overall survival, and disease-free survival.

#### 1.1.3 Exploratory Objective

To determine in some donor recipient pairs the expansion and migration of EBV and CMV-reactive CD8<sup>+</sup> memory T-cells and correlation with EBV and CMV reactivation.

#### 1.2 ClinicalTrials.gov Outcomes

#### 1.2.1 Primary Outcome

**Title**: Graft-versus-Host Disease (GvHD)-free and relapse-free survival (GRFS)

**Description**: The rate of participants who do not experience GvHD and also do not experience relapse are collectively considered to be GRFS. Relapse will be assessed according to the myelodysplastic syndrome or leukemia response criteria. The participants will be assessed for GRFS though 1 year post-transplant. The outcome will be reported as the number of participants, a number without dispersion.

**Timeframe**: 1 year **Safety Outcome?**: No

#### 1.2.2 Secondary Outcomes

Title: Graft Rejection

**Description**: Graft rejection will be determined on the basis of reaction against the donor hematopoietic cells. The outcome will be reported as the number of participants who experience graft rejection though 1 year post-transplant, a number without dispersion.

**Timeframe**: 1 year **Safety Outcome?**: No

**Title**: Acute Graft-versus-Host Disease (GvHD)

**Description**: The participants will be assessed for acute graft-versus-host disease (GvHD) though 1 year post-transplant. The outcome will be reported as the number of participants who experience acute GvHD, a number without dispersion.

**Timeframe**: 1 year **Safety Outcome?**: Yes

**Title**: Chronic Graft-versus-Host Disease (GvHD)

**Description**: The participants will be assessed for chronic, steroid-requiring graft-versus-host disease (GvHD) though 1 year post-transplant. The outcome will be reported as the number of participants who experience chronic GvHD, a number without dispersion.

**Timeframe**: 1 year **Safety Outcome?**: No

**Title**: Non-relapse Mortality

**Description**: Non-relapse mortality will be assessed as the number of participants who have died though 1 year post-transplant, without a relapse or recurrence of their myelodysplastic syndrome or leukemia. Relapse will be assessed according to the myelodysplastic syndrome or leukemia response criteria. The outcome will be reported as the number of affected participants, a number without dispersion.

**Timeframe**: 1 year **Safety Outcome?**: No

Title: Relapse

**Description**: Relapse will be assessed according to the myelodysplastic syndrome or leukemia response criteria. The outcome will be reported as the number of participants who experience relapse though 1 year post-transplant, a number without dispersion.

**Timeframe**: 1 year **Safety Outcome?**: No

Title: Overall Survival (OS)

**Description**: Overall Survival (OS) will be assessed as the number of participants who remain alive at 1 year post-transplant. The outcome will be reported as a number without dispersion.

**Timeframe**: 1 year **Safety Outcome?**: No

#### 2. BACKGROUND

### 2.1 Allogeneic Hematopoietic Cell Transplantation for MDS, Acute Leukemia, and CML

Allogeneic hematopoietic cell transplantation (HCT) is a potentially curative therapy for subjects with high-risk MDS and acute leukemia. Following allogeneic HCT, a significant percentage of subjects with otherwise incurable blood cancers using best of care non-transplantation therapies may achieve long-term disease control and are cured. These patients are characterized by developing donor type hematopoiesis and have complete resolution of all disease-related signs, symptoms, and markers. Generally, patients who undergo allogeneic HCT are doing so as a "last ditch" effort for long-term disease control and possibly cure as best of care non-transplant therapies are unlikely to provide this.

The antitumor activity of allogeneic HCT is from the direct cytotoxic effect of the conditioning regimen combined with the immunologic graft-versus-tumor (GVT) effect mediated by alloreactive donor T-cells. A myeloablative conditioning regimen is the current standard of care for patients with MDS and acute leukemia, as shown in a recent randomized controlled trial demonstrating significantly lower relapse rates and superior overall survival with myeloablative conditioning compared to reduced intensity conditioning (RIC) for fit patients age 18 to 65 with MDS or acute leukemia. <sup>1</sup> The main causes for treatment failure following allogeneic HCT are disease relapse, acute and chronic GvHD, and infections. A strategy to augment donor-mediated GVT activity and improve infection control without increasing the risk of acute and chronic GvHD may improve transplant outcomes including overall survival.

#### 2.2 CD34-Selected Allogeneic HCT for MDS, Acute Leukemia, and CML

CD34 selection with immunomagnetic beads is an effective method of depleting alloreactive donor T-cells from a peripheral blood graft and results in a significant reduction in acute and chronic GvHD. <sup>2-9</sup> Studies of CD34-selected HCT for various hematologic malignancies performed at Memorial Sloan Kettering Cancer Center (MSKCC) reported incidences of acute GvHD (limited to Grade II) of 8%, and chronic GvHD of 9% in recipients of matched related grafts and incidences of acute and chronic GvHD of 9% and 29%, respectively, in recipients of matched unrelated donors. <sup>3,4</sup> None of the subjects received GvHD prophylaxis beyond T-cell depletion of the graft. Results from single-center studies have been validated in the National Blood and Marrow Clinical Trials Network (BMT CTN) study 0303 in which 44 subjects with AML in CR1 or CR2 were conditioned with total body irradiation, thiotepa, and cyclophosphamide with rabbit antithymocyte globulin (ATG) followed by CD34-selected allogeneic HCT from an HLA-matched sibling donor. The incidence of acute GvHD Grade II-IV was 22.7% and the incidence of extensive chronic GvHD was 6.8% at 24 months. <sup>5</sup> Similar results have been reported in subjects with high-risk MDS. In a recent study of 102 subjects at MSKCC with advanced MDS who received CD34-selected HCT, the cumulative incidence of acute GHVD (Grade II to IV) at 180 days was 16% and the cumulative incidence of chronic GvHD at 1 year was 4%. <sup>10</sup> A recent analysis of the BMT CTN 0303 subjects compared to a subset of subjects on BMT CTN 0101 who received a conventional transplant for AML in CR1/CR2 showed a significantly lower rate of chronic GvHD at 2 years with a CD34-selected graft than a conventional graft (19% vs 50%, respectively, p < 0.001, Figure 1) with no difference in overall or disease-free survival. 11



**Figure 1.** Cumulative incidence of chronic GvHD in recipients of CD34-selected T-cell depleted (TCD) grafts compared to recipients of unmanipulated grafts with post-transplant immunosuppressive therapy (IST), Pasquini, *et al*, *J Clin Oncol* 2012.

Another advantage of CD34-selected HCT is that no post-transplant GvHD prophylaxis is required, thus eliminating the risks of side effects like nephrotoxicity associated with calcineurin inhibitors (CNIs) and the combined toxicity of an ablative regimen and methotrexate, which may exacerbate mucositis and cytopenias. The ability to avoid post-transplant immunosuppression also makes CD34-selected HCT an ideal platform for post-transplant adoptive cellular therapies targeting minimal residual disease or infections. <sup>12</sup>

Subject accrual to a multicenter phase 3 trial (BMT CTN 1301, NCT02345850) was recently completed; this trial randomized subjects with MDS or acute leukemia to one of three arms following myeloablative conditioning and transplantation from an HLA-matched donor. Subjects were randomized to either: a CD34-selected graft, an unmanipulated graft followed by post-transplant cyclophosphamide (PTCy), or an unmanipulated graft with conventional post-transplant immunosuppressive therapy consisting of a CNI combined with methotrexate; all three arms are currently accepted standard-of-care approaches for GHVD prophylaxis. The results from the trial may still be more than 18 months from being publically disclosed, albeit interim DSMB analyses throughout has found no evidence of superiority or inferiority in any of the three arm that was sufficient to warrant early closure for safety or efficacy concerns.

#### 2.3 CD34<sup>+</sup> Selection Impact on Disease Relapse, Infection, and Graft Rejection

A major concern limiting the widespread adoption of CD34-selected, T-cell depleted (TCD) donor grafts is loss or attenuation of the GVT effect mediated by alloreactive donor T-cells, which appears to lead to a higher risk of disease relapse. This was first demonstrated in patients with chronic myelogenous leukemia (CML), where a retrospective study of 46 patients who underwent TCD transplants were compared to 40 patients who received conventional grafts. <sup>13</sup>

The 3-year probability of disease relapse was significantly higher in the TCD group than in the non-TCD group (62% vs 24%, p = .0003). The infusion of supplemental donor T-cells was beneficial to the TCD group as after a donor lymphocyte infusion (DLI), 17 of 20 patients in the TCD group and 2 of 3 patients in the non-TCD group achieved a complete remission.

While the CML experience clearly showed a higher risk for disease relapse with a TCD graft, this relationship has not been clearly demonstrated in patients with acute leukemia or MDS. For example, in the BMT CTN 0303 study, the relapse rate for patients with acute leukemia in CR1 receiving a CD34-selected graft was 17.4% at 36 months, similar to historical controls receiving conventional grafts. <sup>5</sup> Another retrospective study compared 115 patients who received TCD grafts after myeloablative conditioning at MSKCC to a cohort of 181 patients who received unmodified grafts after conditioning with busulfan/fludarabine and GvHD prophylaxis with tacrolimus and mini-methotrexate at MD Anderson Cancer Center (MDACC). There were no significant differences in the rate of disease relapse at 3 years between the TCD and unmodified graft recipients (18% vs 25%, p = 0.3). <sup>8</sup> Similarly, in a study of 102 patients with advanced MDS who received CD34-selected grafts at MSKCC, the cumulative incidence of relapse was 11.8% at 1 year and 15.7% at 2 years, <sup>11</sup> similar to historical controls receiving unmodified grafts. The prospective randomized phase 3 BMT CTN 1301 study will be pivotal in comparing CD34-selected HCT to an unmodified graft with either PTCy or standard CNI-based immunosuppression in patients with advanced MDS and acute leukemia.

Another important limitation of CD34-selected TCD grafts is the increased risk for infection, particularly viral reactivation with CMV and EBV, with a higher incidence of EBV-associated lymphoproliferative disorders. <sup>14-18</sup> Prior studies of CD34-selected HCT have demonstrated delayed reconstitution of CD4+ T-cells with a large proportion of patients having absolute CD4+ counts < 200 cells/uL for more than seven months, which may contribute to the increased risk for severe, recurrent, or opportunistic infections. <sup>3</sup>

Early studies of TCD grafts were limited by higher rates of graft rejection than with conventional grafts, with reported graft failure rates as high as 27%. <sup>19-21</sup> These clinical results confirmed pre-clinical data that donor-derived T-cells facilitate engraftment. However, following modification of the conditioning regimen, and in particular the use of ATG to promote engraftment, several centers have reported consistent engraftment with CD34-selected TCD grafts. <sup>2,5,22,23</sup>

# 2.4. CD8<sup>+</sup> Memory T-cells Have GVT Activity Without Causing Severe GvHD in Murine Models of Transplantation

Murine studies showed that in many strain combinations memory T-cells, including memory CD4<sup>+</sup> and memory CD8<sup>+</sup> T-cells induce significantly less GvHD than naïve T-cells (CD62L<sup>hi</sup>CD44<sup>lo</sup>) or combinations of naïve and memory T-cells. <sup>24-30</sup>

Accordingly, our group at Stanford compared isolated naïve CD4+, CD8<sup>+</sup>, or total T-cells, and/or memory CD4+CD44<sup>hi</sup>; CD8<sup>+</sup>CD44<sup>hi</sup>; and total memory CD44<sup>hi</sup> T-cells from unprimed donors for their capacity to induce GvHD, promote chimerism and mediate antitumor activity against a naturally occurring B-cell lymphoma (BCL1) in an MHC-mismatched model. <sup>31</sup> Only the CD8<sup>+</sup>CD44<sup>hi</sup> memory T-cell subset containing both central and effector memory cells was

capable of eradicating the lymphoma cells without inducing GvHD. In contrast, CD4+ and CD8<sup>+</sup> naïve T-cells, memory CD44<sup>hi</sup> CD4+ T-cells, naive total T-cells, and memory CD44<sup>hi</sup> total T-cells either induced lethal GvHD or lacked potent antitumor activity. The tumor-bearing recipients of CD8<sup>+</sup>CD44<sup>hi</sup> T-cells had a clear survival advantage over those given CD8<sup>+</sup> naive T-cells because of the lethal GvHD induced by the latter. The CD8<sup>+</sup>CD44<sup>hi</sup> T-cells were also used in a model of treatment of progressive lymphoma growth after BMT, and were able to promote complete chimerism and eradicate the tumor without causing GvHD.

In other preclinical murine models of bone marrow transplantation using various MCH-matched strain combinations conducted by our group, the only cell subset that we could identify that provided GVT reactions against FBL3 leukemia tumor cells without inducing lethal GvHD was CD44<sup>hi</sup>CD8<sup>+</sup> memory T-cells. <sup>32</sup>

Taken together, our studies and those by other groups suggest that CD8<sup>+</sup> memory T-cells promote donor cell engraftment and retain GVT reactions without precipitating severe GvHD.

#### 2.5 Methods for the Enrichment of Human CD8<sup>+</sup> Memory T-cells

Since we successfully treated progressive tumor growth after BMT without inducing GvHD in mice with purified donor CD8<sup>+</sup> memory T-cells, we developed methods to translate this work to human clinical trials. In studies using healthy donor PBMC apheresis collections and immunomagnetic bead separation on Miltenyi columns, we enriched for CD8<sup>+</sup>CD45RO<sup>+</sup>CD45RA<sup>-</sup> phenotypic memory T-cells to > 95% purity. <sup>33</sup>

Briefly, phenotypic CD8<sup>+</sup> memory T-cells (CD8<sup>+</sup>CD45RA<sup>-</sup>) were isolated from healthy donors following one or two 12-liter volume apheresis collections. The CD45RA<sup>-</sup> cells were obtained by labeling peripheral blood collections with the research grade CliniMACS CD45RA Microbeads (Catalogue number 130-020-003) and Reagent (Miltenyi Biotec) followed by selection on the CliniMACS Plus instrument using program Depletion 3.2 with CliniMACS Depletion tubing sets. The flow through CD45RA<sup>-</sup> cells were labeled with the research grade CliniMACS CD8 Microbeads (Catalogue number 130-030-810) and Reagent and selected using program Enrichment 3.1 with standard CliniMACS tubing sets. Post-selection products were washed and re-suspended in 100 mL of Normosol-R with 1% human serum albumin (HSA) and evaluated immediately and after 24 to 48 hours of storage at 4°C. Products were infused fresh (ie, not cryopreserved) and there was no change in cell viability or phenotype during the 48-hour storage time compared to immediate analysis. Cell viability (consistently > 90%), recovery and purity were determined by flow cytometry, and a representative example is shown in **Figure 2** with > 95% of cells consistent with the CD8<sup>+</sup> memory T-cell subset.



Cell yields were determined using apheresis products from normal HCT donors and the mean  $CD8^+$  memory T-cell post-enrichment cell count obtained from a single 12-liter apheresis product was 8 x  $10^8$  with a range of 5 to 8 x  $10^8$  CD45RA-CD8+ cells. Therefore, following 2 standard volume aphereses or one large volume (18 to 22 liters) apheresis per donor, we estimated that the highest feasible dose of memory  $CD8^+$  T-cells available for infusion would be  $10 \times 10^8$  cells. Assuming that most subjects weigh less than 100 kg, attainable numbers of  $CD8^+$  memory T-cells for a phase 1 dose escalation trial would be  $1 \times 10^6/\text{kg}$ ;  $5 \times 10^6/\text{kg}$ ; and  $10 \times 10^6/\text{kg}$ .

In further studies, the purified phenotypic CD8<sup>+</sup> memory T-cells were tested for immune reactivity *in vitro* by stimulation with irradiated allogeneic PBMCs from normal donors. <sup>33</sup> The responder CD8<sup>+</sup> memory T-cells showed a modest increase in the mean 3H-thymidine incorporation in cultures with allogeneic stimulator cells compared to control cultures without allogeneic stimulators (**Figure 3A**). The CD8<sup>+</sup> memory T-cell supernatants showed a marked increase in the concentration of IFN-γ after culture with allogeneic stimulator cells and a minimal increase in the concentration of IL-2 (**Figure 3B**). The results of the human mixed leukocyte response (MLR) experiments were consistent with the responses observed with CD8<sup>+</sup> memory T-cells from mice where the murine responder cells also showed a modest increase in 3H-thymidine incorporation after stimulation with allogeneic cells, and the production of IFN-γ was considerably greater than that of IL-2.



**Figure 3A.** Proliferation of CI stimulators (Stim) and assessed shown (n = 4). **B.** Cytokine se irradiated allogeneic stimulator Bead Arrays for INF $\gamma$ , IL-2, an

## 2.6 Phase 1 Trial of CDo Intelliory 1 -cell infusion for Kelapseu Hematologic Malignancies after Allogeneic HCT

To test the DLI treatment concept of human donor-derived CD8<sup>+</sup>CD45RO<sup>+</sup>CD45RA<sup>-</sup> memory T-cells in patients, a 15-subject phase 1 safety and feasibility study was conducted under an approved IND (BB-IND-14844) entitled "A Phase I Study of CD8<sup>+</sup>CD45RO<sup>+</sup>CD45RA<sup>-</sup> Memory T-cell Donor Lymphocyte Infusion for Relapse of Hematolymphoid Malignancies Following Matched Related Donor Allogeneic Hematopoietic Cell Transplantation" (NCT01523223). The study followed a standard 3+3 dose escalation format using a low CD8<sup>+</sup> memory T-cell dose of 1 x 10<sup>6</sup> cells/kg, an intermediate dose of 5 x 10<sup>6</sup> cells/kg and a final dose of 10 x 10<sup>6</sup> cells/kg. The objectives of the protocol were:

1. To determine the feasibility of purifying allogeneic CD8<sup>+</sup> memory T-cells suitable for clinical application and to determine the safety and maximum tolerated dose (MTD) of these cells in subjects with recurrent or refractory hematolymphoid malignancies following allogeneic HCT.

- 2. To determine disease response, time to disease progression, event-free survival, and overall survival following treatment with allogeneic CD8<sup>+</sup> memory T-cells.
- 3. To assess donor specific chimerism before and at designated time points after treatment with allogeneic CD8<sup>+</sup> memory T-cells.

Eligible subjects were 18 to 75 years of age. Phenotypic CD8<sup>+</sup> memory T-cells were isolated following 1 or 2 days of unmobilized donor apheresis using a tandem immunomagnetic selection strategy including CD45RA depletion followed by CD8<sup>+</sup> enrichment on the CliniMACS Plus instrument. Fifteen subjects received CD8<sup>+</sup> memory T-cells at 3 dose levels. The subject characteristics and outcomes are summarized in Table 1 and have been previously reported. <sup>34</sup>

Table 1. Subject Outcomes Following CD8<sup>+</sup> Memory T-cell DLI for Disease Relapse after Allogeneic HCT

| Subject | Diagnosis | Disease Status at<br>CD8 <sup>+</sup> Memory<br>Infusion | CD8 <sup>+</sup> Memory Dose (x 10 <sup>6</sup> /kg) | Response<br>following<br>DLI | Time from DLI to<br>Relapse/Progression<br>(Days) | Time from DLI to<br>Death or Last<br>Follow-up (Days) | Status at Last<br>Follow Up |
|---|---|---|---|---|---|---|---|
| 1 | AML | CR2 | 1.0 | CR2 | 973 | 1057 | Expired |
| 2 | AML | Active Disease | 1.0 | CR2 | 480 | 591 | Expired |
| 3 | AML | CR3 | 1.0 | CR3 | 579 | 1328 | Alive in CR |
| 4 | AML | CR2 | 5.0 | CR2 | 120 | 430 | Expired |
| 5 | CML | CR3 | 5.0 | CR3 | - | 1069 | Alive in CR |
| 6 | CLL | Active Disease | 5.0 | PD | NR | 168 | Expired |
| 7 | AML | Active Disease | 7.8 | PD | NR | 128 | Expired |
| 8 | AML | Active Disease | 8.0 | PD | NR | 151 | Expired |
| 9 | NHL | Active Disease | 10.0 | PD | NR | 495 | Alive with disease |
| 10 | NHL | Active Disease | 5.2 | SD | 90 | 412 | Alive with disease |
| 11 | AML | CR2 | 10.0 | CR2 | - | 328 | Alive in CR |
| 12 | AML | CR3 | 7.7 | CR3 | 147 | 286 | Alive with disease |
| 13 | NHL | Active Disease | 10.0 | SD | 158 | 194 | Expired |
| 14 | MM | Active Disease | 10.0 | PD | NR | 221 | Alive with disease |
| 15 | ALL | Active Disease | 10.0 | PR | - | 118 | Alive with disease |

AML, acute myeloid leukemia; CML, chronic myeloid leukemia; CLL, chronic lymphocytic leukemia; NHL, non-Hodgkin lymphoma; MM, multiple myeloma; ALL, acute lymphoblastic leukemia; CR, complete remission; PD, progressive disease; SD, stable disease; PR, partial response; NR, no response

All subjects in dose levels 1 and 2 received the intended  $CD8^+$  memory T-cell dose of 1 to  $10^6$ /kg and 5 to  $10^6$ /kg, respectively. Five of the subjects treated at dose level 3 received the 10 to  $10^6$ /kg  $CD8^+$  memory T-cell dose; however, the intended dose could not be obtained in

4 subjects, who received doses of 5.2 to  $10x10^6$ /kg. The maximum tolerated dose (MTD) was not reached.

No adverse events occurred during CD8<sup>+</sup> memory T-cell infusion, and no dose-limiting toxicities were observed. GvHD developed in only 1 subject, was limited to Grade II involvement of the liver, and resolved following a course of corticosteroids.

Thirteen subjects (87%) received cytoreductive therapy prior to CD8<sup>+</sup> memory T-cell infusion, and 6 subjects (40%) had returned to complete remission (CR) at the time of infusion. The median follow-up from the time of CD8<sup>+</sup> memory T-cell infusion was 328 days (range, 118 to 1328 days). Ten subjects (67%) maintained or achieved an objective response (7 CR; 1 partial response; 2 stable disease) for at least 3 months following CD8<sup>+</sup> memory T-cell infusion, and four of these responders had active disease at time of infusion. Among the 10 responders; 7 have relapsed at the time of this report after a median 165 days (range, 90 to 973 days) to relapse. Eight subjects are currently alive; 3 are alive in CR and 5 are alive with active disease. For the entire study cohort, the median event-free survival and overall survival following CD8<sup>+</sup> memory T-cell infusion were 4.9 months (95% CI, 1 month to 19.3 months) and 19.6 months (95% CI; 5.6 months to not reached), respectively.

In summary, this phase 1 trial showed that CD8<sup>+</sup> memory T-cell DLI is well tolerated and associated with a low incidence of GvHD. The MTD was not reached even at the higher dose level of 10 x 10<sup>6</sup>/kg; however, this yield was unable to be achieved using the current-cell selection strategy. Some subjects achieved a prolonged CR in this small heterogeneous study population with heavily pretreated hematologic malignancies. There did not appear to be a dose response to CD8 memory T-cell infusions as responses were observed at all doses used, and likewise there was not a dose that was associated with increase in toxicity or side effects. Importantly, this clinical trial defined that the dose of phenotypic CD8<sup>+</sup>CD45RO<sup>+</sup>CD45RA<sup>-</sup> T<sub>M</sub> cells reliably obtained for use in a clinical trial using our enrichment strategy is 1 to10 x 10<sup>6</sup>/kg.

# 2.7 Phase 2 Trial of Consolidative CD8<sup>+</sup> Memory T-cell Infusion for Subjects with Mixed Chimerism after Allogeneic HCT

Based on the results of the Phase 1 study that confirmed safety and suggested some level of efficacy, we initiated a second clinical trial entitled "Post-Transplant Infusion of Allogeneic CD8 Memory T-cells as Consolidative Therapy After Non-Myeloablative Allogeneic Hematopoietic Cell Transplantation in Patients with Leukemia and Lymphoma", (NCT02424968) under IND BB-14844. The study rationale is based on multiple publications, including our own, that showed that persistence of mixed hematopoietic cell chimerism after allogeneic HCT was associated with a significantly higher risk of disease relapse. <sup>35-44</sup> Once a patient's disease has relapsed after allogeneic HCT, the ability to return the patient to a durable remission is poor. Therefore, a strategy that can help promote conversion from mixed chimerism (MC) to full donor chimerism (FC) and that does not promote significant GvHD has the potential to improve the outcomes of transplant recipients by reducing the risk of disease relapse.

The primary objective of this study will be to determine the rate of conversion from MC to FC following a post-transplant infusion (day 30 to 70) of enriched donor phenotypic CD8<sup>+</sup> memory T-cells in subjects with hematologic malignancies who received non-myeloablative HCT with

TLI-ATG conditioning. It is hypothesized that subjects who convert from MC to FC will have a reduced risk of relapse similar to subjects who are achieve FC without DLI. The secondary objectives are to determine the risk of disease relapse, overall and event-free survival, non-relapse mortality, and the incidence of acute and chronic GvHD following the infusion of allogeneic CD8<sup>+</sup> memory T-cells.

Eligible subjects are 18 to 75 years of age with a high-risk or refractory hematologic malignancy and who receive nonmyeloablative allogeneic HCT using TLI-ATG conditioning and cells from an HLA-matched donor and who have MC (< 95% donor CD3<sup>+</sup> cells) at day +30. Phenotypic CD8<sup>+</sup> memory T-cells are isolated from HLA-matched donors following 1 or 2 days of apheresis using the tandem immunomagnetic selection strategy including CD45RA depletion followed by CD8<sup>+</sup> enrichment on the CliniMACS Plus instrument. Cell purity is determined by flow cytometry analysis. CD8<sup>+</sup> memory T-cells are planned for infusion between day +30 and day +70 at a dose of 1 to 10 x  $10^6$  cells/kg, the dose determined from the phase 1 trial (Section 2.6, above) to be the maximum dose that can be consistently collected from 1 or 2 apheresis products.

This study will follow a single-arm, Simon 2-stage trial principle. In Simon stage 1, 9 subjects are planned for enrollment, and if three or fewer subjects responded, defined as the conversion from mixed to complete chimerism within 90 days of the CD8<sup>+</sup> T<sub>M</sub> cell infusion, the study will be stopped for futility. If 4 or more subjects respond in Simon stage 1, then in stage 2 enrollment will be planned to continue to a full sample of 18 subjects. Success will be declared if a total of 13 or more subjects respond.

To date, 9 subjects have been enrolled on the trial and received prophylactic donor CD8<sup>+</sup>CD45RO<sup>+</sup>CD45RA<sup>-</sup> memory T-cells between day 30 to 70 post-transplant. <sup>45</sup> Following the CD8<sup>+</sup> memory DLI, subjects were assessed for the development of acute and chronic GvHD, conversion from MC to FC (≥ 95% donor CD3<sup>+</sup> chimerism) within 3 months, and for disease relapse. Secondary outcomes included the incidence of adverse events, invasive infections, non-relapse mortality, overall survival (OS), and disease-free survival (DFS). The subjects and their outcomes are shown in Table 2. <sup>45</sup>

Table 2. Subject characteristics and outcomes following consolidative CD8<sup>+</sup> memory T-cell DLI

| Age/sex | Diagnosis and disease status | | 8 | | 8 | | Day of<br>DLI | pre- and | chimerism<br>d 3 months<br>st-DLI | Acute<br>GvHD | Chronic<br>GvHD | Remission status | Surviving | Follow up<br>days<br>post-HCT |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 71F | AML | CR1 | +40 | 88% | 97% | None | None | CR, MRD negative | Alive | 747 | | | | |
| 67F | AML | CR2 | +33 | 23% | 44% | None | None | Relapsed (day +698) | Alive | 730 | | | | |
| 67M | MDS | PR | +40 | 40% | 19% | None | None | Relapsed (day +88) | Deceased | 128 | | | | |
| 38F | CHL | PR | +42 | 84% | 99% | Grade II<br>(skin) | Mild<br>(joints) | Relapsed (day +231) | Alive | 474 | | | | |
| 47M | DLBCL | PR | +41 | 88% | 95% | None | None | CR | Alive | 390 | | | | |

Table 2. Subject characteristics and outcomes following consolidative CD8<sup>+</sup> memory T-cell DLI

| Age/sex | - C | | Day of pre- and 3 mo DLI post-DLI | | d 3 months | Acute<br>GvHD | Chronic<br>GvHD | Remission status | Surviving | Follow up<br>days<br>post-HCT |
|---|---|---|---|---|---|---|---|---|---|---|
| 60F | DLBCL | CR | +47 | 93% | 100% | Grade II<br>(skin) | None | Relapsed (day +141) | Deceased | 187 |
| 30F | PMBCL | PD | +42 | 88% | 95% | None | None | CR | Alive | 306 |
| 47F | ENKTL | PR | +62 | 75% | 72% | None | None | CR | Alive | 152 |
| 65M | DLBCL | CR | +49 | 92% | 96% | None | None | CR | Alive | 131 |

AML = acute myeloid leukemia; CHL = classical Hodgkin lymphoma; CR = complete remission; DLBCL = diffuse large B-cell lymphoma; DLI = donor lymphocyte infusion; ENKTL = extranodal NK/T-cell lymphoma; GvHD = graft-versus-host disease; HCT = hematopoietic cell transplantation; MDS = myelodysplastic syndrome; MRD = minimal residual disease; PMBCL = primary mediastinal B-cell lymphoma; PD = progressive disease; PR = partial remission

Median age of the subjects was 60 years (range 30 to 71 years) with a median follow up of 306 days post-HCT (range 131 to 747 days). Diagnoses included non-Hodgkin lymphoma (n = 5), AML (n = 2), MDS (n = 1), and Hodgkin lymphoma (n = 1). Median donor CD3<sup>+</sup> chimerism at Day +30 was 88% (range 23 to 93%).

The cell product was highly enriched for  $CD8^+/CD45RA^-/CD45RO^+$  cells, and flow analysis confirmed the selected cells were phenotypically consistent with the  $CD8^+$  T-effector memory subset with a post-enrichment purity of  $\geq 96\%$  (range 96.4 to 98.8%) in all subjects.

CD8<sup>+</sup> memory T-cell DLI was well-tolerated with no adverse events. 6 of the 9 subjects (67%) converted from MC to FC within 3 months post-DLI with a median donor CD3<sup>+</sup> chimerism of 97% (range 95 to 100%). Two subjects developed Grade II acute GvHD (skin only) that was treated to resolution. One subject developed mild chronic GvHD. No subjects developed severe acute GvHD (Grade III to IV) or extensive chronic GvHD. No subjects developed invasive infections, and non-relapse mortality was 0%. Of the 3 subjects who failed to convert from MC to FC, 2 had residual disease at the time of transplant, 1 of whom had early disease relapse at Day +88. 4 of the 6 subjects who converted to FC were in complete remission (CR) at the last follow up. 1 of the 3 subjects with persistent MC was in CR at the last follow up. For the entire study cohort, the median disease-free survival is 1.1 years and the median overall survival is not yet reached.

As with the phase 1 study, the early results from our phase 2 study demonstrate (1) the feasibility of consistently obtaining a cellular product highly enriched for phenotypic CD8<sup>+</sup> memory T-cells at a yield of 1 to 10 x 10<sup>6</sup> cells/kg from donor apheresis products; (2) the safety of this cellular therapy with a very low incidence of mild GvHD and no cases of severe acute GvHD (Grade III-IV) or extensive chronic GvHD observed to date in any of the 24 subjects treated thus far on the phase 1 and phase 2 trials; and (3) the efficacy of CD8<sup>+</sup> memory T-cells in converting 6 of 9 subjects (67%) with MC to FC, recapitulating the results seen in our murine model. Subjects continue to accrue to trial, and further accrual and longer follow up are needed to determine if this strategy will reduce relapse rates for high-risk subjects with MC.

#### **2.8** Proposed Study Rationale and Hypothesis

CD34 selection with immunomagnetic beads is an effective method of depleting alloreactive donor T-cells from a peripheral blood graft, and results in a significant reduction in acute and chronic GvHD. <sup>3,46.47</sup> Yet in these trials, overall subject survival did not appear improved perhaps due to an increase in tumor relapse; graft rejection; and infection. Our **hypothesis** is that combining CD8<sup>+</sup>CD45RA<sup>-</sup> T<sub>M</sub> phenotype cells to a purified CD34<sup>+</sup> graft will retain the low incidence of GvHD, yet also provide protection from graft rejection; protection from infection; and enhance anti-tumor activity compared with CD34<sup>+</sup> selection alone. The proposed trial has particular significance especially in context of the current BMT CTN Phase 3 randomized, multicenter trial (BMT CTN 1301) in which a T-cell depleted (TCD) CD34-selected graft was a SOC arm in subjects with hematologic malignancies undergoing myeloablative conditioning for HCT.

#### 2.9 Study Overview

This single institution, single arm, Simon 2-Stage trial will test the hypothesis that combining donor CD8<sup>+</sup>CD45RA<sup>-</sup> T<sub>M</sub> cells with donor CD34<sup>+</sup> selected grafts will be safe, and that the adoptively transferred CD8<sup>+</sup> T<sub>M</sub> cells into the recipient will enhance anti-tumor, and anti-infection reactions without aggravating GvHD compared with CD34<sup>+</sup> selection alone. **The primary study objective** is the one-year rate of GvHD-free, Relapse-Free Survival (GRFS) as previously defined. <sup>48,49</sup> As with other CD34-selected graft trials, post-transplant immunosuppression will not be used in this trial.

#### 3. PARTICIPANT SELECTION AND ENROLLMENT PROCEDURES

#### 3.1 Eligibility Criteria and Participant Eligibility Checklist

Inclusion and Exclusion Criteria are provided on the Eligibility Checklist, following, and which may be extracted from this document for use in screening potential subjects. otherwise indicated: Pre-transplant screening: all studies to be completed within 70 days of beginning conditioning therapy, unless otherwise indicated:

The Inclusion and Exclusion Criteria are provided on the Participant Eligibility Checklist following, which must be completed in its entirety for each subject prior to registration. The checklist may be extracted from this document for use in screening potential subjects. The completed, signed, and dated checklist must be retained in the subject's study file, and the study's Regulatory Binder.

Pursuant to Stanford Medicine SOP "Confirmation of Participant Eligibility in Clinical Trials," the treating Physician (investigator); the Study Coordinator; and an Independent Reviewer will verify that the subject's eligibility is accurate; complete; and legible in source records. A description of the eligibility verification process should be included in the EPIC or other Electronic Medical Record progress note.

#### **Participant Eligibility Checklist**

#### I. Protocol Information

| Protocol Title: | CD34-Selected Allogeneic Hematopoietic Cell Transplantation with Myeloablative Conditioning and CD8 <sup>+</sup> Memory T-cell Infusion For Patients with Myelodysplastic Syndrome, Acute Leukemia, and Chronic Myelogenous Leukemia (CML) |
|---|---|
| eProtocol number:<br>OnCore number: | |
| Principal Investigator: | Robert Lowsky, MD |

#### II. Subject Information

| Subject name / Unique ID: | | / |
|---------------------------|--------|--------|
| Gender | ☐ Male | Female |

#### III. Eligibility Criteria

#### **RECIPIENT Inclusion Criteria**

Pre-transplant screening: all studies to be completed within 70 days of beginning conditioning therapy, unless otherwise indicated.

| Prospective RECIPIENTS Must MATCH ALL these Inclusion Criteria to be Eligible | Yes | No | Supporting Documentation * |
|---|---|---|---|
| Acute leukemia, in morphologic complete remission; <b>OR</b> myelodysplasia with < 10% blasts in the marrow, and no circulating blasts that contain auer rods; <b>OR</b> chronic myelogenous leukemia (CML) with any one of the following high-risk features: | | | |
| 1. Chronic Phase CML yet with additional karyotypic features at diagnosis that are beyond the reciprocal translocation (9;22)(q34;q11) known as Philadelphia (Ph) chromosome. | | | |
| 2. Resistant CML, defined as: | | | |
| <ul> <li>A failure of therapy to achieve a complete<br/>cytogenetic response within 12 months of<br/>diagnosis,</li> </ul> | | | |
| <ul> <li>A failure of therapy to maintain a &gt; 3 log-fold<br/>reduction in molecular response once beyond<br/>12 months of treatment,</li> </ul> | | | |
| <ul> <li>Any new leukemia-associated<br/>chromosomal/sequence abnormality detected by<br/>conventional cytogenetics; FISH; molecular or<br/>next generation sequencing.</li> </ul> | | | |
| • Enlarging spleen size despite ongoing treatment. | | | |
| 3. Accelerated Phase CML, defined as: | | | |
| • 10% to 19% blasts in the blood and/or bone marrow. | | | |
| <ul> <li>&gt; 20% basophils in the peripheral blood.</li> </ul> | | | |
| <ul> <li>Any new leukemia-associated<br/>chromosomal/sequence abnormality detected by<br/>conventional cytogenetics; FISH; molecular or<br/>next generation sequencing.</li> </ul> | | | |
| 4. Blast Crises CML, defined as: | | | |
| • > 20% marrow or blood blasts. | | | |
| Subjects with chronic myelomonocytic leukemia (CMML) must have a WBC count $\leq$ 10,000 cells/ $\mu$ L and $<$ 10% blasts in the marrow. | | | |
| Planned myeloablative conditioning regimen at<br>Stanford University Medical Center. | | | |

| Prospective RECIPIENTS Must MATCH<br>ALL these Inclusion Criteria to be Eligible | Yes | No | Supporting Documentation * |
|---|---|---|---|
| 2. ≥ 18 years to < 66.0 years | | | |
| 3. Males or females | | | |
| 4. Karnofsky or Lansky Performance Score ≥ 70%. | | | |
| 5. Must have an HLA-matched donor as follows: donor must be an 8/8 match for HLA-A, -B and -C at intermediate (or higher) resolution, and -DRB1 at high resolution using DNA-based typing. The donors must be willing to receive G-CSF followed by collection of cells by apheresis, and must meet the Program's criteria for donation. | | | |
| 6. Cardiac function: Ejection fraction at rest ≥ 40% | | | |
| 7. Serum creatinine value of < 1.5 mg/dL, or an estimated creatinine clearance greater than 50 mL/minute (using the Stanford calculator for eGFR available in EPIC) | | | |
| 8. Diffusing capacity of the lungs for carbon monoxide (DLCO) ≥ 50% (adjusted for Hgb) | | | |
| 9. Forced vital capacity (FVC) ≥ 50% | | | |
| 10. Forced expiratory volume (FEV1) ≥ 50% | | | |
| 11. Total bilirubin < 2 times the upper limit of normal (ULN) (unless the elevated bilirubin is attributed to Gilbert's Syndrome) | | | |
| 12. Alanine aminotransferase (ALT) < 2.5 x ULN | | | |
| 13. Aspartate aminotransferase (AST) < 2.5 x ULN | | | _ |
| 14. Signed informed consent | | | |

#### **RECIPIENT Exclusion Criteria**

| Prospective RECIPIENTS Must <u>NOT</u> Match<br><u>ANY</u> of These Exclusion Criteria | Yes | No | Supporting Documentation * |
|---|---|---|---|
| Prior autologous or allogeneic hematopoietic stem cell transplant | | | |
| 2. Prior malignancies, except resected non-melanoma or treated cervical carcinoma <i>in situ</i> . Cancer treated with curative intent ≥ 5 years previously is allowed. Cancer treated with curative intent < 5 years previously will not be allowed unless approved by the Protocol Officer or one of the Protocol Chairs | | | |
| 3. Active CNS involvement by malignant cells | | | |
| 4. Presence of fluid collection (ascites, pleural or pericardial effusion) that interferes with methotrexate clearance or makes methotrexate use contraindicated | | | |
| 5. Requirement for supplemental oxygen | | | |
| 6. Uncontrolled bacterial, viral or fungal infections (currently taking medication and with progression or no clinical improvement) at time of enrollment | | | |
| 7. History of uncontrolled autoimmune disease or on active treatment (defined as > 5 mg prednisone daily) | | | |
| 8. Seropositive for HIV-1 or -2 | | | |
| 9. Seropositive for HTLV-I or –II | | | |
| 10. Active Hepatitis B or C viral replication by PCR | | | |
| 11. Documented allergy to iron dextran or murine proteins | | | |

| Prospective RECIPIENTS Must <u>NOT</u> Match<br><u>ANY</u> of These Exclusion Criteria | Yes | No | Supporting Documentation * |
|---|---|---|---|
| 12. Pregnant (positive serum or urine βHCG) or breastfeeding) | | | |
| 13. Females of childbearing potential (FCBP) or men who have sexual contact with FCBP unwilling to use an effective form of birth control or abstinence for one year after transplantation | | | |
| 14. Unable to comply with the treatment protocol, including appropriate supportive care, follow-up and research tests | | | |
| 15. Planned to receive post-transplant maintenance therapy except for FLT3 inhibitors or BCR-ABL tyrosine kinase inhibitors (TKIs) | | | |
| * All subject files must include supporting documentation method of confirmation can include, but is not limited to, results, subject self-report, and medical record review. | | | |
| V. Statement of Eligibility (RECIPIENT) By signing this form of this trial I verify that this subject is: eligible / ineligible for participation in the study. This study is approved by the Stanford Cancer Institute Scientific Review Committee, the IRB of record, and has finalized financial and contractual agreements as required by Stanford School of Medicine's Research Management Group. | | | |
| Study Coordinator printed name: | | | Date: |
| Signature: | | | |
| | | | D. |
| Investigator printed name: Date: | | | |
| Signature: | | | |
| Triple-check reviewer printed name: | | | Date: |
| Signature: | | | |

| Trottocor ritie. | Myeloablative Conditioning and Patients with Myelodysplastic Syl Chronic myelogenous leukemia ( | CD8 <sup>+</sup> N<br>ndrom | <b>1emo</b> | ry T-cell Infusion For |
|---|---|---|---|---|
| eProtocol number:<br>OnCore number: | IRB-49023<br>BMT339 | | | |
| Principal Investigator: | Robert Lowsky, MD | | | |
| DONOR name / Uniq | ue ID: | | / | |
| Gender | Gender | | | |
| | iteria - Donors for this trial will follow<br>nobilized hematopoietic cell donors at | _ | | |
| | DONOR Must MATCH<br>Ision Criteria to be Eligible | Yes | No | Supporting Documentation * |
| 1. HLA-matched donor (matching at 8/8 antigens or alleles including HLA-A, -B, -C, and –DRB1). | | | | |
| 2. ≥ 18 years to < 66.0 years | | | | |
| 3. State of general good health | | | | |
| 4. Completed a donor evaluation with history, medical examination and standard blood tests within 60 days of starting the hematopoietic cell collection procedure. In order to fairly represent the interests of the donor, the donor evaluation and consent will be performed by a study team member other than the recipient's attending physician. | | | | |
| 5. Hepatitis A, B and C, HIV-1 and -2, HTLV, VZV, EBV, HSV, West Nile virus, Syphilis Treponema, T cruzi (Chagas), CMV, and the MPX NAT IDT (HIV/HCV/HBV) will be tested as per national standard of care guidelines for transplant donors. Donors who are HIV-positive will be excluded. Donors who are positive by serology for Hepatitis B or C are eligible as long as PCR for RNA/DNA is negative | | | | |
| 6. White blood cell count > $3.5 \times 10^9$ /L | | | | |

| Prospective DONOR Must MATCH ALL these Inclusion Criteria to be Eligible | | No | Supporting Documentation * |
|---|---|---|---|
| 7. Platelets > $150 \times 10^9 / L$ | | | |
| 8. Hematocrit > 35% | | | |
| 9. Capable of undergoing leukapheresis | | | |
| 10. Able to understand and sign informed consent | | | |
| DONOR Exclusion Criteria | | | |
| Prospective DONOR Must <u>NOT</u> Match <u>ANY</u> of These Exclusion Criteria | Ye<br>s | No | Supporting Documentation * |
| Psychological traits or psychological or medical conditions which make them unlikely to tolerate the procedure | | | |
| 2. Pregnant or lactating female | | | |
| * All subject files must include supporting documentation to confirm subject eligibility. The method of confirmation can include, but is not limited to, laboratory test results, radiology test results, subject self-report, and medical record review. | | | |
| V. Statement of Eligibility (DONOR) | | | |
| By signing this form of this trial I verify that this subject is: eligible / ineligible for participation in the study. This study is approved by the Stanford Cancer Institute Scientific Review Committee, the IRB of record, and has finalized financial and contractual agreements as required by Stanford School of Medicine's Research Management Group. | | | |
| Study Coordinator printed name: | | | Date: |
| Signature: | | | |
| Investigator printed name: | | | Date: |
| Signature: | | | |
| Triple-check reviewer printed name: | | ] | Date: |
| Signature: | | | |

#### 3.2 Recruitment and Informed Consent

Subjects will be selected based upon the eligibility requirements highlighted above. Informed consent forms will be approved by the Stanford University IRB, SRC and FDA. No payment will be provided to participate in this protocol. Costs for routine care will be borne by the subject's insurance carrier. Research costs including cell enrichment procedures of the CD8<sup>+</sup> T<sub>M</sub> cells as well as all research studies will be borne by an NCI-sponsored Program Project Grant (PPG 4P01CA049605-27).

#### 3.3 Potential Risk to the Recipient

Subjects who undergo allogeneic HCT have risks for a variety of complications that include transplant-related deaths. An Attending Physician will explain the risks associated with HCT in detail to the subject and their caregivers once it is deemed that treatment with this protocol is a feasible consideration and appropriate. The physician involved in the consenting process will not be the primary physician who is involved in managing the care of the subject or donor. A detailed discussion regarding the current alternative treatment which is a CD34-selected graft without a CD8<sup>+</sup> memory T-cell infusion, an unmanipulated donor graft with SOC post-transplant immune suppression or post-transplant Cyclophosphamide will be discussed with the subject and their caregiver(s). All inclusion criteria eligibility must be fulfilled. The plan will also be discussed with the subject's referring physician.

Potential Sensitization to Murine Proteins: Mouse protein antibodies are used in the CliniMACS processing procedures. If the recipient has a pre-existing allergy, he or she may be at risk for allergic reactions during infusion of the processed cells; although the residual amount of murine protein in the final product is very low (estimated maximum dose for a 50 kg subject would be  $30~\mu g$ ). To date, no allergic reactions are reported in subjects receiving cells processed with the CliniMACS System. Epinephrine and antihistamines will be available at the recipient's bedside during the PBSC infusion.

#### 3.4 Protection Against Risks

The patient-subject will receive a consent form with appropriate information concerning the cell infusion. Risks include the toxicities of the acute and chronic GvHD, infection, marrow aplasia and cytopenia, disease progression, and the possible other unforeseen risks given the novel nature of the clinical trial. All questions will be answered by the Attending Physician as well as Nurse Coordinator. The physician involved in this process will not be the primary physician who is involved in managing the care of the patient-subject or donor. Once a patient-subject has agreed to proceed with the trial a formal 1 to 1.5 hour consenting process will be performed by the Research Nurse and all questions will be answered. Signed informed consent must be obtained prior to initiation of the protocol. Risks to the donors are expected to be very low and are the same as for other donors who undergo collection for traditional HCT.

To maintain confidentiality, study subject identification will not be revealed in any reports or publications resulting from the study. Information will be provided to the study subjects' physicians as necessary, to the IRB, DSMB, and FDA as necessary. Case report forms and other study records will not identify the subjects by name. To monitor data and safety of the research, the procedures as outlined in the "Data and Safety Monitoring Plan" (see below) will be followed.

#### 3.5 Potential Benefits of the Proposed Research to the Subjects

This study represents a logical extension of our work on the use of CD8<sup>+</sup> T<sub>M</sub> cells that have the potential to improve transplant outcomes by providing anti-tumor activity and enhancing post-transplant immune reconstitution with prevention from infection yet without increasing the risk of GvHD. The potential benefits could be realized by patient-subjects who participate in this trial, yet it is understood that the trial concept and design is investigational.

#### 3.6 Importance of the Knowledge to be Gained

The goal of the trial is to test the treatment concept that adding HLA matched donor CD8<sup>+</sup>CD45RA<sup>-</sup> T<sub>M</sub> phenotype cells to purified CD34<sup>+</sup> grafts given to recipients undergoing full dose conditioning and HCT for acute leukemia and MDS is safe, and will reduce the risk of disease relapse and infections without increasing the risk of GvHD. If we are successful, it is likely that this strategy will improve overall subject survival. As well, the strategy developed in the proposed trial can be effectively adapted to other clinical transplant settings, and therefore has applicability to treat diseases beyond acute leukemia and MDS. The overall significance is a potential improvement in transplant outcomes.

#### 3.8 Inclusion of Women and Minorities

Women and minorities and are eligible for this protocol.

#### 3.9 Subject Withdrawal

Participation in the trial is voluntary. Subjects will be advised that they may voluntarily withdraw from the study at any time and will be instructed to notify the investigator. Subjects may choose to withdraw for any reason(s). Subjects are not obligated to reveal their reason(s) for withdrawal to the sponsor.

#### 3.10 Subject Withdrawal from Data Collection

If a subject explicitly states they do not wish to contribute further data to the trial their decision must be respected and notified to the sponsor in writing. In this event details should be recorded in the subject's hospital records, no further CRFs must be completed and no further data sent to the sponsor.

#### 4 TREATMENT PLAN

#### **Study Transplant Conditioning Regimen**

#### **OPTION 1:**

Fractionated TBI will be delivered in the standardized format consisting of a total dose of 1375 cGy given in fractions on days -10 -9,-8 and -7. Sequential doses are administered in an anterior/posterior or lateral orientation. The orientation of TBI chosen will be left to the discretion of the radiation oncologist but will remain consistent at our institution throughout the duration of the trial. Full value lung blocks are not used yet compensators and lung blocks yielding a minimum of 800 cGy lung dose are allowed based on our institutional practice. Depending on the method of lung shielding employed, the blocked areas should be boosted with high-energy electrons or be otherwise radiated so that the cumulative chest wall dose is approximately 1300 cGy, so as to ensure that marrow sites in the ribs are adequately treated. In

addition, male subjects receiving transplants for ALL or AML, use of boost to testes is allowed according to institutional practices.

**Thiotepa** will be administered at 5 mg/kg/day intravenously over 4 hours for 2 consecutive days (Day -6 and -5).

**Fludarabine** will be administered intravenously over 30 minutes at a total dose of 125 mg/m<sup>2</sup> divided into 5 daily doses of 25 mg/m<sup>2</sup>/day (Day -6 to -2).

#### **Treatment Schedule**

| Days -10 to -7 | Fractionated TBI | (1375 cGy), | , administered over 4 days |
|----------------|------------------|-------------|----------------------------|
|----------------|------------------|-------------|----------------------------|

Days -6 to -5 Thiotepa 5 mg/kg/day: IV for 2 consecutive days

Days -6 to -2 Fludarabine 25 mg/m<sup>2</sup>/day: IV for 5 consecutive days

#### **OPTION 2: : Non TBI Conditioning – Busulfan/Cyclophosphamide**

- Days -7 to -4: Busulfan: 3.6 mg/kg/dose Q24h IV. Infused over 3 hours. 1 dose per day x 4 consecutive days x 3.6 mg/kg/dose = 14.4 mg/kg
- Days -3 to -2 Cyclophosphamide: 60 mg/kg/dose Q24h IV. Infused over 2 hours. 1 dose per day x 2 consecutive days x 60 mg/kg/dose = 120 mg/kg

#### **Immune Suppression Medication**

Tacrolimus .01 mg/kg IV BID or .03 mg/kg PO BID

- 1. Begin day -3
- 2. Target serum level is 5-10 ng/ml
- 3. If > 15 kg over IBW, dose based on adjusted IBW

Dose adjusted based on creatinine, t. bilirubin and serum drug levels.

Tacrolimus taper will begin around day +90 in the absence of GVHD and based on clinical decisions. The aim will be to discontinue Tacrolimus altogether if clinically applicable (no history of GVHD) by around day +180. In some patients who are considered higher risk for disease relapse, as determined by the medical team, the tacrolimus taper may begin in the absence of active GVHD by day +60.

#### 4.2 Hematopoietic Stem Cell Graft Collection

Transplant donors are considered research subjects by the FDA. For HLA-matched donors, the consent process will be done at the Stanford University Medical Center along with routine donor consent procedures according to institutional guidelines. The donor informed consent document for donors will be reviewed and approved by the Stanford University IRB.

#### 4.3 Mobilization of Donor

Following screening and enrollment, donors will undergo 1 to 2 days of apheresis collections for the processing and enrichment for CD34+ cells and for CD8+CD45RA-  $T_M$  cells as detailed in Section 5. As per standard of care, donor mobilization will be using G-CSF (filgrastim or its biosimilar equivalent) and cell collection will be done using standard procedures for apheresis. A sample donor schedule is described below, and as per standard of care the schedule can shift one day up or down depending on apheresis and CTF (cell therapy facility) availability. In general, the donor will begin GCSF on Day -6 or Day -7 of the conditioning regimen at a dose of  $10 \,\mu g/kg/day$  actual body weight subcutaneously (rounded to a multiple of the nearest vial size of either 300 or 480  $\mu g$ ). Based on the volume of GCSF, the dose may be split into multiple injection sites. The mobilization phase will start on the  $1^{st}$  day of administration of G-CSF (Day -6 or Day -7) and continue until the final day of leukapheresis (Day -1 or Day -2). The donor will undergo their  $1^{st}$  apheresis on Day -2 or Day -3, and if it is determined that an additional apheresis is required to achieve adequate cell doses, then a  $2^{nd}$  apheresis will be on Day -1 or Day -2, respectively. Therefore, the cell collection days for the donor will be Days -3 and -2, or it can be Days -2 and -1.

#### 4.3 Donor Leukapheresis

Leukapheresis will be performed on a continuous flow cell separator according to institutional standards and will commence on the morning of the fifth day of G-CSF treatment. The anti-coagulant used for the procedure will be acid citrate dextrose (ACD). The volume of blood processed per leukapheresis session should be approximately three to four times total blood volume as tolerated by the donor. It is expected that many donors will undergo 2 consecutive days of apheresis. Concurrent plasma (about 200 mLs) will be collected for products to be stored overnight. A unique identification and labeling system will be used to track the leukapheresis product from collection to infusion according to FACT/JACIE guidelines.

#### 5 INVESTIGATIONAL AGENT INFORMATION

#### 5.1 Investigational Agent: CD8<sup>+</sup> Memory T-Cell Selection

The apheresis product will be enriched for CD8<sup>+</sup>CD45RA<sup>-</sup> memory T-cells. In a procedure we successfully used in 2 prior clinical trials, we will enrich for donor CD8<sup>+</sup> memory T-cells using a tandem immunomagnetic selection procedure that involves the CliniMACS Cell Selection System (Miltenyi Biotec). Depletion of CD45RA expressing cells uses CliniMACS CD45RA Reagent (BB-MF-11872). The CD45RA depleted fraction is then enriched for CD8-expressing cells by positive cell selection with CliniMACS CD8 Reagent (BB-MF-11704). The cells will be infused in the usual manner on Day 0 and within 6 hours of the CD34<sup>+</sup> selected stem cell infusion.

In our two prior clinical trials we determined that 2 consecutive days of aphereses per donor will yield a target cell dose of 5 to  $10 \times 10^6 \, \text{CD8}^+$  memory T-cells/kg for all subjects, assuming most subjects weigh less than  $120 \, \text{kg}$ . We will use a dose range of 5 to  $10 \times 10^6 \, \text{CD8}^+$  memory T-cells/kg for the current study, as both dose levels ( $5 \times 10^6 \, \text{kg}$  and  $10 \times 10^6 \, \text{kg}$ ) were well tolerated in our prior phase 1 study. We will not exceed a dose of  $10 \times 10^6 \, \text{CD8}^+$  memory T-cells/kg. If the number of CD8<sup>+</sup> memory T-cells falls below the desired threshold of

 $5 \times 10^6$ /kg, the infusion will proceed as planned because we believe it is in the subject's best interest to receive the cell infusion. The CD8<sup>+</sup> memory T-cell infusion has the potential to help achieve donor cell engraftment, provide anti-tumor reactions and protect from infections yet without increasing the GvHD risk. It is expected that a cell yield of  $< 5 \times 10^6$ /kg will be obtained less than 20% of the time.

#### 5.2 Stability

As part of our original IND, we submitted stability data to the FDA from validation runs that extended to 72 hours from the time of completion of first apheresis, and showed negligible loss in cell viability as all validation products continued with > 90% viability. In addition, the results from our prior CD8<sup>+</sup> memory T-cells trials confirmed stability data extending to 72 hours after completion of first apheresis from 8 additional donors, and all cases maintained > 94% viability.

#### 5.3 Reagents for cells for immediate release and conditions for storage

The CD8 and CD45 reagent systems are pharmaceutical grade and both have Master Files that are BB-MF-11704 and BB-MF-11872, respectively. Donors will undergo two consecutive apheresis days with the first day of apheresis being in the afternoon expected to begin around 2 PM and be completed by 6 PM (the collection will be stored overnight in a 4-degree Celsius bio-fridge), followed by a second apheresis the next morning starting at around 7:30 AM. The two days of collections will be batched for routine SOC CD34<sup>+</sup> cell selection that will be performed on the same day as the second collection. The CD34<sup>+</sup> flow through will be diluted for overnight storage at 4 degrees Celsius with 1 volume of Normosol-R with 2% HSA. Thereafter, the following morning the tandem immunomagnetic selection procedure for enrichment of CD45RA<sup>-</sup>CD8<sup>+</sup> phenotype T-cells will be performed. For subject comfort, the final volume of the infusate will be reduced to < or equal to 200 mL and the CD8<sup>+</sup> memory T-cell concentration will range between 1 x 10<sup>6</sup> to 1 x 10<sup>8</sup> cells/mL. The final infusate will be diluted in the Miltenyi Biotech Selection Buffers that contain PBS with 1mmolar EDTA and 0.5% HSA. It is estimated that all CD45RA-CD8<sup>+</sup> phenotype T-cell products will be infused within 72 hours from completion of the first apheresis.

#### 5.4 Release Requirements of the Product

Release of the selected cell products for infusion includes:

- Negative Gram staining (no organisms detected).
- Endotoxin levels  $\leq 0.5$  EU/milliliter of infused product volume
- 80% cell viability as assessed by trypan blue or 7-AAD dye exclusion.
- $\geq$  80% of the CD3+ cells express the CD8 memory T-cell phenotype, here defined as:
  - $\circ$  CD8<sup>+</sup>/CD45RA<sup>-</sup>/CD45RO<sup>+</sup>
  - $\circ \le 5\%$  of cells with the CD3<sup>+</sup>/CD45RA<sup>+</sup>/CD45RO<sup>-</sup> phenotype
  - $\circ$  Sufficient cells with the CD8 memory T-cell phenotype to meet the desired dose, or at least the minimum dose of  $> 2 \times 10^6$  CD8<sup>+</sup> memory T-cells/kg

In addition, post-selection sterility cultures in accordance with sterility testing guidelines (21CFR§610.12) will be conducted to confirm the sterility of the selected cells. Any positive growth results obtained will be documented in the processing record of the selection and immediately communicated to the subject's attending physician in accordance with the plan of action for the infusion of cellular products with microbial contamination. Ancillary studies may include phenotypic analysis of the selected cells and cytokine secretion profiles from MLR assays may be used to further our understanding of the CD8<sup>+</sup> memory T-cell population characteristics but do not constitute release criteria at this time. If the cell product does not meet release criteria after manipulation, the product will not be infused.

In the case(s) where the manipulated cell product does not meet release criteria, the subject will be removed from the study due to a failure to receive the investigational product. If 2 of the first 5 enrolled subjects fail to receive the CD8<sup>+</sup> memory T-cell product due to a failure to satisfy the release criteria, a formal DSMC review will be initiated. An enrolled subject who does not receive the CD8<sup>+</sup> memory T-cell product will be removed from the study and replaced with another subject as the accrual target is 30 subjects who will be infused with CD8<sup>+</sup> memory T-cells.

#### **6 DOSE MODIFICATION**

As a single treatment transplant procedure, dose modification for any particular subject is not anticipated.

#### 7 ADVERSE EVENTS AND REPORTING PROCEDURES

#### 7.1 Adverse Events

Hematopoietic cell transplantation (HCT) is an aggressive therapy for the treatment of a number of life-threatening disorders, including cancer. In this setting, a very large number of Grade 1, 2 and 3 adverse events (AEs) are expected to occur, regardless of whether or not a subject is participating in a research study. In order to minimize the "background noise" and to focus on clinically significant, meaningful adverse events useful in the assessment of proposed trial the following AE reporting schema is proposed. This schema is intended to capture all AEs that are clinically significant and/or impactful, but minimize "not informative" AE collection.

Laboratory values without a clinical consequence or outcome will not be recorded as adverse events, unless deemed serious (see below).

Grade 1 to 3 AEs not meeting these criteria will not be collected, except as follows. Grade 1 to 3 AEs resulting in subject termination or withdrawal from the study will be collected.

An adverse event is considered a serious adverse event (SAE) if it fulfills one of the following SAE criteria per 21CFR§312.32(a):

- Results in death.
- Life-threatening (subject at risk of death at the time of the event).
- Requiring new inpatient hospitalization or prolongation of existing hospitalization.
- Resulting in persistent or significant disability.
- Other medical events that may not be immediately life-threatening or result in death or hospitalization by may jeopardize the subject or require intervention to prevent one of the outcomes listed above

Grade 4 and higher AEs will be collected and documented with causality attribution on an adverse event log (AE log), and all AEs meeting the criteria of "serious" as defined at 21CFR§312.32(a), including any that are otherwise Grade 1, 2 or 3 will be collected; identified as serious; and documented on an AE log, including causality attribution.

All SAEs will be collected as outlined in Section 7.1 from date of CD8<sup>+</sup> memory T-cell infusion through 365 days. All SAEs will be tracked until resolution or at least 60 days after the study treatment.

Vital signs for all subjects enrolled on the trial will be monitored for infusion-related toxicities (AEs) during the CD8 memory T-cell infusion, and every 30 minutes for 2 hours afterwards. Observed events will be recorded on the AE log. In particular, subjects will be observed for hemodynamic instability, allergic reactions (eg, hives, rashes, angioedema), and fevers (> 38.3°).

The development of acute GvHD, its date of onset and overall grade, is a key secondary outcome measure for subjects on this trial. Acute GvHD will be recorded on an AE log.

#### 7.2 Adverse Event Reporting

All SAEs will be reported to the IRB; to the IND; and to the DSMC, either in an annual review or as an expedited report, in accordance with the established practices of the Stanford Division of Blood and Marrow Transplantation, as well as applicable guidelines and regulations. AEs meeting the criteria specified for an IND Safety Report as defined at 21CFR§312.32(c)(1) will be collected; documented in the adverse event log; and reported to the IND (on a MedWatch 3500A form) in the timeframe specified. The IND annual report will include summaries of the collected AEs, as specified by 21CFR§312.33.

#### 8 CORRELATIVE/SPECIAL STUDIES

None planned.

#### 9 STUDY CALENDAR

| | Pre-Enrollment requirements <sup>A</sup> | On-study enrollment <sup>A</sup> = CD8 <sup>+</sup><br>Memory T-cell Infusion (Day 0) | Time (days) from on-study enrollment ± 20 days | | • |
|---|---|---|---|---|---|
| | | | Day +90 | <b>Day 180</b> | <b>Day 365</b> |
| CD34 <sup>+</sup> cell Infusion | | X | | | |
| Infusion of CD8 <sup>+</sup> memory<br>T-cells | | X | | | |
| Informed consent | X | | | | |
| Demographics | X | | | | |
| Medical history | X | | X | X | X |
| Donor evaluation | X | | | | |
| Physical exam | X | | X | X | X |
| Fulfills inclusion criteria | X | | | | X |
| Has no exclusion criteria | X | | | | |

| Performance status | X | X | X | X |
|---------------------------------------------------------|---|---|---|---|
| Disease Status<br>Assessment | X | X | X | X |
| CBC with differential | | X | X | X |
| Serum chemistry | | X | X | X |
| STR analysis <sup>B</sup> | | X | X | X |
| Assess for ≥ Grade 2 acute GvHD <sup>C</sup> | | X | X | X |
| Assess for moderate or severe chronic GvHD <sup>C</sup> | | X | X | X |

All pre-transplant screening and procedures must be completed within 70 days of beginning conditioning therapy (unless otherwise indicated).

B STR analysis will only be performed beyond Day +90 if there is concern about mixed chimerism or relapse.

Refers to if the event was recorded during the reporting periods of Day 0 to +90; Day 91 to +180; and Day 181 to +365.

#### 10. MEASUREMENTS

#### 10.1 Primary and Secondary Objectives and Outcome measures

Objectives and outcome measures are described at Section 1.1 and 1.2.

#### 11. REGULATORY CONSIDERATIONS

#### 11.1 Institutional Review of Protocol

The protocol, the proposed informed consent and all forms of participant information related to the study (eg, advertisements used to recruit participants) will be reviewed and approved by the Stanford IRB and Stanford Cancer Institute Scientific Review Committee (SRC). Any changes made to the protocol will be submitted as a modification and will be approved by the IRB prior to implementation. The Protocol Director will disseminate the protocol amendment information to all participating investigators.

#### 11.2 Data and Safety Monitoring Plan

The Stanford Cancer Institute Data and Safety Monitoring Committee (DSMC) will be the monitoring entity for this study. The DSMC will audit study-related activities to determine whether the study has been conducted in accordance with the protocol, local standard operating procedures, FDA regulations, and Good Clinical Practice (GCP). This may include review of the following types of documents participating in the study: regulatory binders, case report forms, eligibility checklists, and source documents. In addition, the DSMC will regularly review serious adverse events and protocol deviations associated with the research to ensure the protection of human subjects. Results of the DSMC audit will be communicated to the IRB and the appropriate regulatory authorities at the time of continuing review, or in an expedited fashion, as needed.

#### 11.3 Data Management Plan

The Protocol Director, or his/her designee, will prepare and maintain adequate and accurate participant case histories with observations and data pertinent to the study, in accordance with the established practices of the Stanford Division of Blood and Marrow Transplantation. Accrual rates will be reported to the Data Safety Monitoring Committee (DSMC) and data quality will be reviewed by the Study Statistician. The DSMC of the Stanford Cancer Center will oversee this study and will receive regular reporting of SAEs and monitoring. This Committee involves knowledgeable physicians, scientists and statisticians who oversee all phase I/II trials conducted under the auspices of the Stanford Cancer Center. Individuals who serve on this Committee who are associated with this trial will recuse themselves from discussions of study results, and decisions about revision or closure. Audits will be conducted as requested. Data will also be submitted to the FDA as required by our IND and follow the appropriate reporting rules and regulations including an annual report.

#### 11.4 Good Clinical Practice Guidelines

The clinical investigators assure that the clinical study is performed in accordance with the protocol, the ICH Harmonized Tripartite Guidelines for Good Clinical Practice 1996, the Declaration of Helsinki (Recommendations guiding physicians in Biomedical Research involving Human Subjects; Helsinki 1964; and as amended Tokyo 1975; Venice 1983;

Hong Kong 1989; Somerset West 1996; Edinburgh 2000; Seoul 2008; and Fortaleza 2013) and applicable regulatory requirements.

#### 12. STATISTICAL CONSIDERATIONS

#### 12.1 Statistical Design

The study is a single arm, Simon 2-stage trial with a modification to avoid protracted temporary closure of accrual at the end of the first stage. In single and multi-center studies consisting of over 1500 adult patients treated with SOC allogeneic HCT, the 1-year probability of GRFS was 30%. <sup>48,49</sup> For Type 1 and 2 error rates of 0.10 and 0.2 respectively (power of 0.80), a control success rate of 0.30 and experimental rate of 0.50, the Simon optimal design calls for enrolling 15 subjects in stage 1 and if 6 or more subjects achieve success, then in stage 2 continuing to enroll to a full sample of 32 subjects and declare success if a total of 13 subjects experience success. In order to avoid a protracted temporary closure between the first and second stage, Day 100 GRFS will be evaluated at the 1<sup>st</sup> stage. If  $\geq$  6 subjects in Simon stage 1 are alive without relapse or Grade III-IV GvHD at Day +100, then the full cohort of 32 subjects will be enrolled for stage 2. Success will be declared if  $\geq 13$  subjects of 32 meet the primary endpoint of GRFS at 1 year, and if at least 6 of the stage 1 subjects ultimately meet that endpoint as well. With that proviso, this modified design has the same type 1 and 2 errors of a hypothetical standard Simon 2-stage design which would pause at the end of stage 1 until at least 6 subjects reach the 1-year GRFS outcome. However, the modification modestly increases the expected number of subjects treated (under the null, as discussed below).

Note that the end of stage 1 is defined as 100 days, while at the final analysis is for 1 year. Subjects who fail at 100 days will be regarded as failing in the time frame of the final analysis. No increase in type I or type II error is anticipated.

#### 12.1.1 Randomization

This is a single arm, non-randomized study.

#### 12.2 Interim analyses

There is no formal plan for an interim analysis because the intrinsic nature of the Simon two-stage design is such that the study will not proceed to stage 2, unless the null hypothesis is rejected, because activation of the second stage depends on an adequate number of success observed in the first stage. Therefore, the trial design incorporates stopping early for futility and safety. It is possible that CD8<sup>+</sup>CD45RA<sup>-</sup> T<sub>M</sub> cells will induce acute GvHD. If 2 of the first 4 subjects develop Grade 2 or higher acute GvHD, or, if after 8 subjects, > 30% develop Grade 2 or higher acute GvHD, then we will include a post-transplant GvHD prophylactic regimen. Toxicity, adverse events, and other safety endpoints will be monitored regularly and reported to the DSMB at each meeting or earlier. The expected 100-day mortality rate for a myeloablative transplant is 15 to 20% based on our data as well as CIBMTR data. The rate of mortality will be monitored up to 100 days after transplant, and if 2 of the first 4 enrolled subjects, or if 3 subjects in Simon stage one die within 100 days of transplant, this will trigger a DSMB safety review. If 2 subjects experience graft rejection in Simon stage one, this too will trigger a DSMB review.

#### 12.3 Primary endpoint

The primary endpoint is GvHD-free, relapse-free survival (GRFS) at 1 year. Development of acute GvHD Grade 3 or higher, extensive chronic GvHD requiring immunosuppression, relapse, or death will be considered failures for this endpoint.

#### 12.4 Sample Size

#### 12.4.1 Accrual estimates

32 subjects is the full target accrual for the study.

#### 12.4.2 Sample size justification

It is estimated that 1 subject per month will be accrued. The total subject accrual is expected to take approximately 32 months. Given that accrual rate, the 15<sup>th</sup> (last) subject recruited for stage 1 will reach the +100 day milestone at about 18 months of study time, and the first 6 subjects recruited will have reached the 1-year point. The entire first stage group of 15 subjects will reach the 1-year milestone at month 27. Thus, sometime between the end of months 18 and 27, it will be known whether the unmodified Simon trial would be stopped. During that interim period, up to 9 new subjects would be recruited. This is an upper bound on the excess exposure under the null. It is approached only if the +100 day GRFS rate is considerably larger than the 1-year GRFS rate null, so that few of the first-stage +100 day successes continue to 1 year. We have no direct estimate of the failure rate over 1 year given GRFS at +100 days (under the experimental treatment), so we do not attempt to refine the calculation further.

#### 13. REFERENCES

- 1. Scott BL, Pasquini MC, Logan BR, *et al.* Myeloablative Versus Reduced-Intensity Hematopoietic Cell Transplantation for Acute Myeloid Leukemia and Myelodysplastic Syndromes. *J Clin Oncol*. 2017;35(11):1154-1161.
- 2. Papadopoulos EB, Carabasi MH, Castro-Malaspina H, *et al.* T-cell-depleted allogeneic bone marrow transplantation as postremission therapy for acute myelogenous leukemia: freedom from relapse in the absence of graft-versus-host disease. *Blood.* 1998;91(3):1083-1090.
- 3. Jakubowski AA, Small TN, Young JW, *et al.* T-cell depleted stem-cell transplantation for adults with hematologic malignancies: sustained engraftment of HLA-matched related donor grafts without the use of antithymocyte globulin. *Blood.* 2007;110(13):4552-4559.
- 4. Jakubowski AA, Small TN, Kernan NA, *et al.* T-cell-Depleted Unrelated Donor Stem Cell Transplantation Provides Favorable Disease-Free Survival for Adults with Hematologic Malignancies. *Biol Blood Marrow Transplant.* 2011.
- 5. Devine SM, Carter S, Soiffer RJ, *et al.* Low risk of chronic graft-versus-host disease and relapse associated with T-cell-depleted peripheral blood stem cell transplantation for acute myelogenous leukemia in first remission: results of the blood and marrow transplant clinical trials network protocol 0303. *Biol Blood Marrow Transplant.* 2011;17(9):1343-1351.
- 6. Castro-Malaspina H, Jabubowski AA, Papadopoulos EB, *et al.* Transplantation in remission improves the disease-free survival of patients with advanced myelodysplastic syndromes treated with myeloablative T-cell-depleted stem cell transplants from HLA-identical siblings. *Biol Blood Marrow Transplant*. 2008;14(4):458-4568.
- 7. Perales MA, Jenq R, Goldberg JD, *et al.* Second-line age-adjusted International Prognostic Index in patients with advanced non-Hodgkin lymphoma after T-cell depleted allogeneic hematopoietic SCT. *Bone Marrow Transplant.* 2010;45(9):1408-1416.
- 8. Goldberg JD, Linker A, Kuk D, *et al.* T-cell-Depleted Stem Cell Transplantation for Adults with High-Risk Acute Lymphoblastic Leukemia: Long-Term Survival for Patients in First Complete Remission with a Decreased Risk of Graft-versus-Host Disease. *Biol Blood Marrow Transplant.* 2013;19(2):208-213.
- 9. Bayraktar UD, de Lima M, Saliba RM, *et al.* Ex Vivo T-cell Depleted versus Unmodified Allografts in Patients with Acute Myeloid Leukemia in First Complete Remission. *Biol Blood Marrow Transplant.* 2013.
- 10. Tamari R, Chung S, Papdopoulos EB, *et al.* CD34-selected hematopoietic stem cell transplants conditioned with myeloablative regimens and anti-thymocyte globulin for advanced myelodysplastic syndrome: limited graft-versus-host disease without increased relapse. *Biol Blood Marrow Transplant.* 2015;21(12):2106-2114.
- 11. Pasquini MC, Devine S, Mendizabal A, *et al.* Comparative outcomes of donor graft CD34<sup>+</sup> selection and immune suppressive therapy as graft-versus-host disease prophylaxis for patients with acute myeloid leukemia in complete remission undergoing HLA-matched sibling allogeneic hematopoietic cell transplantation. *J Clin Oncol.* 2012;30(26):3194-3201.
- 12. O'Reilly RJ, Koehne G, Hasan AN, *et al.* T-cell depleted allogeneic hematopoietic cell transplants as a platform for adoptive therapy with leukemia selective or virus-specific T-cells. *Bone Marrow Transplant*. 2015;50:S43-50.
- 13. Sehn LH, Alyea EP, Weller E, *et al.* Comparative outcomes of T-cell depleted and non-T-cell-depleted allogeneic bone marrow transplantation for chronic myelogenous leukemia: impact of donor lymphocyte infusion. *J Clin Oncol.* 1999;17(2):561-568.
- 14. Engelhard D, Or R, Strauss N, *et al.* Cytomegalovirus infection and disease after T-cell depleted allogeneic bone marrow transplantation for malignant hematologic diseases. *Transplant Proc* 1989;21:3101-3102.
- 15. Hertenstein B, Hampl W, Bunjes D, *et al.* In vivo/ex vivo T-cell depletion for GvHD prophylaxis influences onset and course of active cytomegalovirus infection and disease after BMT. *Bone Marrow Transplant*. 1995;15:387-393.

- 16. Couriel D, Canosa J, Engler H, *et al*. Early reactivation of cytomegalovirus and high risk of interstitial pneumonitis following T-depleted BMT for adults with hematological malignancies. *Bone Marrow Transplant*. 1996;18: 347-353.
- 17. Zutter MM, Martin PJ, Sale GE, *et al.* Epstein-Barr virus lymphoproliferation after bone marrow transplantation. *Blood.* 1988;72:520-529.
- 18. Shapiro RS, McClain K, Frizzera G, *et al.* Epstein-Barr virus associated B cell lymphoproliferative disorders following bone marrow transplantation. *Blood.* 1988;71:1234-1243.
- 19. Martin PJ, Hansen JA, Buckner CD, *et al.* Effects of in vitro depletion of T-cells in HLA-identical allogeneic marrow grafts. *Blood.* 1985;66(3):664-672.
- 20. Martin PJ, Hansen JA, Torok-Storb B, *et al.* Effects of treating marrow with a CD3-specific immunotoxin for prevention of acute graft-versus-host disease. *Bone Marrow Transplant*. 1988;3(5):437-444.
- 21. Young JW, Papadopoulos EB, Cunningham I, *et al.* T-cell-depleted allogeneic bone marrow transplantation in adults with acute nonlymphocytic leukemia in first remission. *Blood.* 1992;79(12):3380-3387.
- 22. Aversa F, Terenzi A, Carotti A, *et al.* Improved outcome with T-cell-depleted bone marrow transplantation for acute leukemia. *J Clin Oncol.* 1999;17(5):1545-1550.
- 23. Alyea EP, Weller E, Fisher DC, *et al.* Comparable outcome with T-cell-depleted unrelated-donor versus related-donor allogeneic bone marrow transplantation. *Biol Blood Marrow Transplant.* 2002;8(11):601-607.
- 24. Anderson BE, McNiff J, Yan J, *et al.* Memory CD4+ T-cells do not induce graft-versus-host disease. *J Clin Invest.* 2003;112(1):101-108.
- 25. Dutt S, Tseng D, Ermann J, *et al.* Naive and Memory T-cells Induce Different Types of Graft-versus-Host Disease. *J Immunol.* 2007;179(10):6547-6554.
- 26. Zheng H, Matte-Martone C, Li H, *et al.* Effector memory CD4+ T-cells mediate graft-versus-leukemia without inducing graft-versus-host disease. *Blood.* 2008;111(4):2476-2484.
- 27. Zhang Y, Joe G, Zhu J, *et al.* Dendritic cell-activated CD44<sup>hi</sup>CD8<sup>+</sup> T-cells are defective in mediating acute graft-versus-host disease but retain graft-versus-leukemia activity. *Blood.* 2004;103(10):3970-3978.
- 28. Chen BJ, Cui X, Sempowski, *et al.* Transfer of allogeneic CD62L<sup>-</sup> memory T-cells without graft-versus-host disease. *Blood.* 2004. 103(4):1534-1541.
- 29. Chen BJ, Deoliveira D, Cui X, *et al.* Inability of memory T-cells to induce graft-versus-host disease is a result of an abortive alloresponse. *Blood.* 2007;109(7):3115-3123.
- 30. Zheng H, Matte-Martone C, Jain D, *et al*. Central Memory CD8<sup>+</sup> T-cells Induce Graft-versus-Host Disease and Mediate Graft-versus-Leukemia. *J Immunol*. 2009;182(10):5938-5948.
- 31. Dutt S, Baker J, Kohrt HE, *et al.* CD8<sup>+</sup>CD44(hi) but not CD4+CD44(hi) memory T-cells mediate potent graft antilymphoma activity without GvHD. *Blood.* 2011;117(11):3230-9.
- 32. Kohrt HE, Muller A, Baker J, *et al.* Donor immunization with WT1 peptide augments anti-leukemic activity after MHC-matched bone marrow transplantation. *Blood.* 2011;118(19):5319-5329.
- 33. Armstrong R, *et al.* Immunomagnetic Selection of CD8<sup>+</sup> Memory Cells for Therapeutic Applications. *Biol Blood Marrow Transplant*. 2011. 17(2,Supplement 1):S220.
- 34. Muffly LS, Sheehan K, Armstrong R, *et al.* Infusion of donor-derived CD8<sup>+</sup> memory T-cells for relapse following allogeneic hematopoietic cell transplantation. *Blood Adv.* 2018;2(6):681-690.
- 35. Kohrt HE, Turnbull BB, Heydari K, *et al.* TLI and ATG conditioning with low risk of graft-versus-host disease retains antitumor reactions after allogeneic hematopoietic cell transplantation from related and unrelated donors. *Blood.* 2009;114(5):1099-1109.
- 36. Childs R, Clave E, Contentin N, *et al.* Engraftment kinetics after nonmyeloablative allogeneic peripheral blood stem cell transplantation: full donor T-cell chimerism precedes alloimmune responses. *Blood*. 1999;94(9):3234-3241.

- 37. Reshef R, Hexner EO, Loren AW, *et al.* Early donor chimerism levels predict relapse and survival after allogeneic stem cell transplantation with reduced-intensity conditioning. *Biol Blood Marrow Transplant*. 2014;20(11):1758-1766.
- 38. Koreth J, Kim HT, Nikiforow S, *et al.* Donor chimerism early after reduced-intensity conditioning hematopoietic stem cell transplantation predicts relapse and survival. *Biol Blood Marrow Transplant*. 2014;20(10):1516-1521.
- 39. Solomon SR, Sizemore CA, Zhang X, *et al.* Preemptive DLI without withdrawal of immunosuppression to promote complete donor T-cell chimerism results in favorable outcomes for high-risk older recipients of alemtuzumab-containing reduced-intensity unrelated donor allogeneic transplant: a prospective phase II trial. *Bone Marrow Transplant.* 2014;49(5):616-621.
- 40. Rujkijyanont P, Morris C, Kang G, *et al*. Risk-adapted donor lymphocyte infusion based on chimerism and donor source in pediatric leukemia. *Blood Cancer J*. 2013;3:e137.
- 41. Dey BR, McAfee S, Colby C, *et al.* Impact of prophylactic donor leukocyte infusions on mixed chimerism, graft-versus-host disease, and antitumor response in patients with advanced hematologic malignancies treated with nonmyeloablative conditioning and allogeneic bone marrow transplantation. *Biol Blood Marrow Transplant*. 2003;9(5):320-329.
- 42. El-Cheikh J, Crocchiolo R, Furst S, *et al.* Donor CD3(+) lymphocyte infusion after reduced intensity conditioning allogeneic stem cell transplantation: single-center experience. *Exp Hematol.* 2013;41(1):17-27.
- 43. Liga M, Triantafyllou E, Tiniakou M, *et al*. High alloreactivity of low-dose prophylactic donor lymphocyte infusion in patients with acute leukemia undergoing allogeneic hematopoietic cell transplantation with an alemtuzumab-containing conditioning regimen. *Biol Blood Marrow Transplant*. 2013;19(1):75-81.
- 44. Bloor AJ, Thomson K, Chowdhry N, *et al*. High response rate to donor lymphocyte infusion after allogeneic stem cell transplantation for indolent non-Hodgkin lymphoma. *Biol Blood Marrow Transplant*. 2008;14(1):50-58.
- 45. Spinner MA, Muffly LS, Arai S, *et al.* Consolidative CD8<sup>+</sup> Memory T-cell Donor Lymphocyte Infusion Augments Donor Chimerism with a Low Risk of GvHD Following Matched Related Donor Hematopoietic Cell Transplantation. *Blood.* 2017;130:2003.
- 46. Barba P, Hilden P, Devlin SM, *et al.* Ex Vivo CD34<sup>+</sup>-Selected T-cell-Depleted Peripheral Blood Stem Cell Grafts for Allogeneic Hematopoietic Stem Cell Transplantation in Acute Leukemia and Myelodysplastic Syndrome Is Associated with Low Incidence of Acute and Chronic Graft-versus-Host Disease and High Treatment Response. *Biol Blood Marrow Transplant*. 2017;23(3):452-458.
- 47. Devine SM, Carter S, Soiffer RJ, *et al.* Low risk of chronic graft-versus-host disease and relapse associated with T-cell-depleted peripheral blood stem cell transplantation for acute myelogenous leukemia in first remission: results of the blood and marrow transplant clinical trials network protocol 0303. *Biol Blood Marrow Transplant.* 2011;17(9):1343-1351.
- 48. Holtan SG, DeFor TE, Lazrayan A, *et al.* Composite end point of graft-versus-host disease-free, relapse-free survival after allogeneic hematopoietic cell transplantation. *Blood.* 2015;125(8):1333-1338.
- 49. Solomon SR, Sizemore C, Zhang X, *et al.* Current Graft-versus-Host Disease-Free, Relapse-Free Survival: A Dynamic Endpoint to Better Define Efficacy after Allogenic Transplant. Biol Blood Marrow Transplant. 2017;23(7):1208-1214.
- 50. (Bu/Mel/Flu) Conditioning Versus Total Body Irradiation/Thiotepa/Cyclophosphamide (HFTBI/Thio/Cy) Based Conditioning in Patients with Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS) Undergoing CD34-Selected T-Cell Depleted Allogeneic Stem Cell Transplantation (alloSCT). Orozco J., et la. Biol Blood and Marrow Transplant (BBMT): 339: vol 25, Issue 3, March 2019 S276-277.

#### **APPENDICES**

#### APPENDIX A GVHD SCORING CRITERIA

#### Glucksberg clinical stage and grade of acute GvHD

| Stage | Skin | Liver | Intestinal tract |
|---|---|---|---|
| 1 | Maculopapular rash < 25% of body surface | Bilirubin 34–50 μmol/l | > 500 ml diarrhoea/d |
| 2 | Maculopapular rash 25-50% body surface | Bilirubin 51–102 μmol/l | > 1000 ml diarrhoea/d |
| 3 | Generalized erythroderma | Bilirubin 103-225 µmol/l | > 1500 ml diarrhoea/d |
| 4 | Generalized erythroderma with bullous formation and desquamation | Bilirubin > 255 $\mu$ mol/l | Severe abdominal pain<br>with or without ileus |
| Grade | Degree of organ involvement | | |
| Grade<br>I | Degree of organ involvement Stage 1–2 skin rash; no gut involvement; no liver involvement | t; no decrease in clinical perforn | nance |
| Grade<br>I<br>II | | | |
| Grade<br>I<br>II | Stage 1–2 skin rash; no gut involvement; no liver involvemen | nvolvement (or both); mild decre | ease in clinical performan |

#### NIH consensus criteria for chronic GvHD severity with examples

(comprehensive organ scoring criteria is reviewed in Jagasia, et al, BBMT 2014)

| Mild | <ul> <li>1 or 2 organs or sites (except lung) with score 1</li> <li>Mild oral symptoms, no decrease in oral intake</li> <li>Mild dry eyes, lubricant eyedrops ≤ 3x/day</li> </ul> |
|---|---|
| Moderate | <ul> <li>3 or more organs with score 1</li> <li>At least 1 organ or site with score 2 <ul> <li>19-50% body surface area involved or superficial sclerosis</li> <li>Moderate dry eyes, eyedrops &gt; 3x/day or punctal plugs</li> </ul> </li> <li>Lung score 1 (FEV1 60-79% or dyspnea with stairs)</li> </ul> |
| Severe | <ul> <li>At least 1 organ or site with score 3</li> <li>&gt; 50% body surface area involved</li> <li>Deep sclerosis, impaired mobility or ulceration</li> <li>Severe oral symptoms with major limitation in oral intake</li> <li>Severe dry eyes affecting ADL</li> <li>Lung score 2 (FEV1 40-59% or dyspnea walking on flat ground)</li> </ul> |

#### APPENDIX B. RESPONSE CRITERIA by DISEASE HISTOLOGY

AML Response Criteria (Dohner, et al, Blood 2017)

Table 6. Response criteria in AML

| Category | Definition | Comment |
|---|---|---|
| Response | | |
| CR without minimal residual disease (CR <sub>MRD</sub> ) | If studied pretreatment, CR with negativity for a genetic marker by RT-qPCR, or CR with negativity by MFC | Sensitivities vary by marker tested, and by method used; therefore, test used and sensitivity of the assay should be reported; analyses should be done in experienced laboratories (centralized diagnostics) |
| Complete remission (CR) | Bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; $ANC \ge 1.0 \times 10^9 / L \; (1000/\mu L); \; platelet \; count \ge 100 \times 10^9 / L \; (100000/\mu L)$ | MRD <sup>+</sup> or unknown |
| CR with incomplete<br>hematologic recovery<br>(CR <sub>i</sub> ) | All CR criteria except for residual neutropenia ( $<1.0 \times 10^9/L$ [ $1000/\mu L$ ]) or thrombocytopenia ( $<100 \times 10^9/L$ [ $100\ 000/\mu L$ ]) | |
| Morphologic leukemia-free state (MLFS) | Bone marrow blasts <5%; absence of blasts with Auer rods;<br>absence of extramedullary disease; no hematologic recovery<br>required | Marrow should not merely be "aplastic"; at least 200 cells should be enumerated or cellularity should be at least 10% |
| Partial remission (PR) | All hematologic criteria of CR; decrease of bone marrow blast percentage to 5% to 25%; and decrease of pretreatment bone marrow blast percentage by at least 50% | Especially important in the context of phase 1-2 clinical trials |
| Treatment failure | | |
| Primary refractory disease | No CR or CR <sub>i</sub> after 2 courses of intensive induction treatment;<br>excluding patients with death in aplasia or death due to<br>indeterminate cause | Regimens containing higher doses of cytarabine (see Table 8) are generally considered as the best option for patients not responding to a first cycle of 7+3; the likelihood of responding to such regimens is lower after failure of a first |
| Death in aplasia | Deaths occurring ≥7 d following completion of initial treatment while cytopenic; with an aplastic or hypoplastic bone marrow obtained within 7 d of death, without evidence of persistent leukemia | |
| Death from indeterminate cause | Deaths occurring before completion of therapy, or <7 d following its completion; or deaths occurring ≥7 d following completion of initial therapy with no blasts in the blood, but no bone marrow examination available | |
| Response criteria for clinical trials only | | |
| Stable disease | Absence of $CR_{MRD-}$ , $CR$ , $CR_{i}$ , $PR$ , $MLFS$ ; and criteria for PD not met | Period of stable disease should last at least 3 mo |
| Progressive disease (PD)*,† | Evidence for an increase in bone marrow blast percentage and/or increase of absolute blast counts in the blood: | Category mainly applies for older patient given low-<br>intensity or single-agent "targeted therapies" in<br>clinical trials |
| | <ul> <li>&gt;50% increase in marrow blasts over baseline (a minimum 15% point increase is required in cases with &lt;30% blasts at baseline; or persistent marrow blast percentage of &gt;70% over at least 3 mo; without at least a 100% improvement in ANC to an absolute level (&gt;0.5 × 10<sup>9</sup>/L [500/μL], and/or platelet count to &gt;50 × 10<sup>9</sup>/L [50 000/μL] nontransfused); or</li> <li>&gt;50% increase in peripheral blasts (WBC × % blasts) to &gt;25 × 10<sup>9</sup>/L (&gt;25 000/μL) (in the absence of differentiation syndrome)†; or</li> <li>New extramedullary disease</li> </ul> | In general, at least 2 cycles of a novel agent should be administered Some protocols may require blast increase in 2 consecutive marrow assessments at least 4 wk apart; the date of progression should then be defined as of the first observation date Some protocols may allow transient addition of hydroxyurea to lower blast counts "Progressive disease" is usually accompanied by a decline in ANC and platelets and increased transfusion requirement and decline in performance status or increase in symptoms |
| Relapse | | |
| Hematologic relapse | Bone marrow blasts ≥5%; or reappearance of blasts in the | |
| (after CR <sub>MRD</sub> , CR, CR <sub>i</sub> ) | blood; or development of extramedullary disease | Test soulled constitute of the |
| Molecular relapse<br>(after CR <sub>MRD</sub> ) | If studied pretreatment, reoccurrence of MRD as assessed by RT-qPCR or by MFC | Test applied, sensitivity of the assay, and cutoff values used must be reported; analyses should be done in experienced laboratories (centralized diagnostics) |

IRB-49023 Page 42 of 43 12 February 2021 v4

#### ALL Response Criteria (Brown, et al, JNCCN 2017)

#### Response Criteria for Blood and Bone Marrow:

- CR
- ▶ No circulating blasts or extramedullary disease
  - ♦ No lymphadenopathy, splenomegaly, skin/gum infiltration/testicular mass/CNS involvement
- ▶ Trilineage hematopoiesis (TLH) and <5% blasts
- ▶ Absolute neutrophil count (ANC) >1000/microL
- ▶ Platelets >100,000/microL
- No recurrence for 4 weeks
- CR with incomplete blood count recovery (CRi)
- ▶ Meets all criteria for CR except platelet count and/or ANC
- Overall response rate (ORR = CR + CRi)
- Refractory disease
- Failure to achieve CR at the end of induction
- Progressive disease (PD)
- Increase of at least 25% in the absolute number of circulating or bone marrow blasts or development of extramedullary disease
- Relapsed disease
- Reappearance of blasts in the blood or bone marrow (>5%) or in any extramedullary site after a CR

#### MDS Response Criteria (Cheson, et al, Blood 2006)

Table 3. Proposed modified International Working Group response criteria for altering natural history of MDS7

| Category | Response criteria (responses must last at least 4 wk) |
|---|---|
| Complete remission | Bone marrow: $\leq$ 5% myeloblasts with normal maturation of all cell lines* Persistent dysplasia will be noted*† Peripheral blood‡ Hgb $\geq$ 11 g/dL Platelets $\geq$ 100 $\times$ 10 $^9$ /L Neutrophils $\geq$ 1.0 $\times$ 10 $^9$ /L† Blasts 0% |
| Partial remission | All CR criteria if abnormal before treatment except: Bone marrow blasts decreased by ≥ 50% over pretreatment but still > 5% Cellularity and morphology not relevant |
| Marrow CR† | Bone marrow: $\leq$ 5% myeloblasts and decrease by $\geq$ 50% over pretreatment†<br>Peripheral blood: if HI responses, they will be noted in addition to marrow CR† |
| Stable disease | Failure to achieve at least PR, but no evidence of progression for $>$ 8 wks |
| Failure | Death during treatment or disease progression characterized by worsening of cytopenias, increase in percentage of bone marrow blasts, or progression to a more advanced MDS FAB subtype than pretreatment |
| Relapse after CR or PR | At least 1 of the following: Return to pretreatment bone marrow blast percentage Decrement of $\geq 50\%$ from maximum remission/response levels in granulocytes or platelets Reduction in Hgb concentration by $\geq 1.5$ g/dL or transfusion dependence |
| Cytogenetic response | Complete Disappearance of the chromosomal abnormality without appearance of new ones Partial At least 50% reduction of the chromosomal abnormality |
| Disease progression | For patients with: Less than 5% blasts: ≥ 50% increase in blasts to > 5% blasts 5%-10% blasts: ≥ 50% increase to > 10% blasts 10%-20% blasts: ≥ 50% increase to > 20% blasts 20%-30% blasts: ≥ 50% increase to > 30% blasts Any of the following: At least 50% decrement from maximum remission/response in granulocytes or platelets Reduction in Hgb by ≥ 2 g/dL Transfusion dependence |
| Survival | Endpoints: Overall: death from any cause Event free: failure or death from any cause PFS: disease progression or death from MDS DFS: time to relapse Cause-specific death: death related to MDS |